CLINICAL TRIAL: NCT00712933
Title: A Multi-Center, Continuation Trial of Belimumab (HGS1006, LymphoStat-B™)a Fully Human Monoclonal Anti-BLyS Antibody in Subjects With Systemic Lupus Erythematosus (SLE) Who Completed the Phase 3 Protocol HGS1006-C1056 or HGS1006-C1057
Brief Title: A Continuation Trial for Subjects With Lupus That Completed Protocol HGS1006-C1056 or HGS1006-C1057
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112234; 2007-007648-85 (EudraCT Number)
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Belimumab; Antibodies; Systemic Lupus Erythematosus; Lupus; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 1 mg/kg dose of belimumab given IV every 28 days.
  Interventions: Drug: belimumab
- 2. (Experimental): 10 mg/kg dose of belimumab given IV every 28 days.
  Interventions: Drug: belimumab

INTERVENTIONS:
Drug: belimumab — Recombinant, fully human, monoclonal antibody
  Comparison of the 1 mg/kg and 10 mg/kg dose of belimumab given IV every 28 days.
  Other Names: LymphoStat-B™; HGS1006

SUMMARY:
This is a long-term continuation study to provide continuing treatment to subjects with SLE.

DETAILED DESCRIPTION:
This trial is a long-term continuation study to provide continuing treatment to subjects with System Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Have completed the HGS 1006-C1056 or HGS 1006-C1057 protocol through the Week 72 or Week 48 visits, respectively.

Exclusion Criteria:

* Have developed any other medical disease or condition that has made the patient unsuitable for this study in the opinion of their physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2008-05-30 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (92):
- Argentina (6):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
- GSK Investigational Site, Vienna, Austria
- GSK Investigational Site, Liège, Belgium
- Brazil (9):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Goiânia, Goiás
  - GSK Investigational Site, Juiz de Fora, Minas Gerais
  - GSK Investigational Site, Recife, Pernambuco
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago
- Colombia (4):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
  - GSK Investigational Site, Medellín
- Czechia (4):
  - GSK Investigational Site, Brno-Bohunice
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- GSK Investigational Site, Suresnes, France
- Germany (9):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Kiel
- Hong Kong (2):
  - GSK Investigational Site, Chai Wan
  - GSK Investigational Site, New Territories
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Trivandrum
- Israel (5):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
- GSK Investigational Site, Roma, Italy
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, México
  - GSK Investigational Site, San Luis Potosí City
- Netherlands (2):
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
- Peru (3):
  - GSK Investigational Site, Surco, Lima region
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- Philippines (6):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Sampaloc Manila
- GSK Investigational Site, Gmina Końskie, Poland
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Piešťany, Slovakia
- South Korea (6):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- GSK Investigational Site, Stockholm, Sweden
- Taiwan (6):
  - GSK Investigational Site, Dalin Township, Chiayi County
  - GSK Investigational Site, Gueishan Township,Taoyuan County
  - GSK Investigational Site, Hualien City
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20055

REFERENCES:
- [Background] Bruce IN, Urowitz M, van Vollenhoven R, Aranow C, Fettiplace J, Oldham M, Wilson B, Molta C, Roth D, Gordon D. Long-term organ damage accrual and safety in patients with SLE treated with belimumab plus standard of care. Lupus. 2016 Jun;25(7):699-709. doi: 10.1177/0961203315625119. Epub 2016 Mar 1. PMID 26936891
- [Background] van Vollenhoven RF, Navarra SV, Levy RA, Thomas M, Heath A, Lustine T, Adamkovic A, Fettiplace J, Wang ML, Ji B, Roth D. Long-term safety and limited organ damage in patients with systemic lupus erythematosus treated with belimumab: a Phase III study extension. Rheumatology (Oxford). 2020 Feb 1;59(2):281-291. doi: 10.1093/rheumatology/kez279. PMID 31302695
- [Derived] Urowitz MB, Ohsfeldt RL, Wielage RC, Dever JJ, Zakerifar M, Asukai Y, Ramachandran S, Joshi AV. Comparative analysis of long-term organ damage in patients with systemic lupus erythematosus using belimumab versus standard therapy: a post hoc longitudinal study. Lupus Sci Med. 2020 Oct;7(1):e000412. doi: 10.1136/lupus-2020-000412. PMID 33051264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, continuation trial of belimumab and was conducted at 115 centers in 28 countries. Participants with Systemic Lupus Erythematosus (SLE), who had completed the Phase 3 HGS1006-C1056 or HGS1006-C1057 trial or participants who had previously received subcutaneous belimumab in Protocol HGS1006-C1070 were included in this trial.
Pre-assignment Details: 738 participants were enrolled in the study and 735 received at least one dose of belimumab.Out of 735 participants, 368 completed the study and 370 withdrew from the study.
Groups:
- Belimumab 10mg/kg IV: Participants received belimumab every 28 days by intravenous (IV) infusion at 1 milligram per kilogram (mg/kg) or 10 mg/kg body weight. Participants who received either 1 mg/kg or 10 mg/kg belimumab in their parent studies continued to receive the same dose of belimumab. Participants randomized to receive placebo in the parent studies received 10 mg/kg beliumamb. Subsequently, the dose of belimumab for participants receiving 1 mg/kg was increased to 10 mg/kg .All participants also received SoC SLE therapy while participating in this trial.
Period: Overall Study
Arm/Group | Belimumab 10mg/kg IV
Started | 735
Completed | 368
Not Completed | 367
Not completed — Adverse Event | 69
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 22
Not completed — Non-compliance with study drug | 13
Not completed — Other Pregnancy | 37
Not completed — Sponsor decision | 14
Not completed — Withdrew consent | 4
Not completed — Hip replacement surgery | 1
Not completed — Involved in Clinical research | 3
Not completed — Participant hospitalized | 1
Not completed — Participant travelled overseas | 2
Not completed — Death of patient | 1
Not completed — Other Physician decision | 1
Not completed — Not committed to contraception | 1
Not completed — Participant received medication | 1
Not completed — Physician Decision | 36
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 151

BASELINE CHARACTERISTICS:
Population: Modified Intention to Treat (MITT) includes all participants who were enrolled in BEL112234 and were treated with at least one dose of belimumab in the continuation study.
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 695
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American/African Heritage | 18
  American Indian or Alaska Native | 225
  East Asian Heritage | 118
  South Asian Heritage | 38
  Southeast Asian Heritage | 58
  Middle East/North African Heritage | 22
  White/Caucasian/European Heritage | 256

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: An adverse event is defined as any unfavorable or unintended sign, symptom, or disease that is temporally associated with the use of a study agent but is not necessarily caused by the study agent. This includes worsening (example: increase in frequency or severity) of preexisting conditions. Participants with incidences of any event at any time post-baseline are presented by yearly interval. Only treatment-emergent AEs are summarized.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Participants
  Any-time post Baseline,n=735 | 706
  Year 0-1,n=735 | 617
  Year 1-2 ,n =701: number analyzed (Participants) | 701
  Year 1-2 ,n =701 | 502
  Year 2-3, n= 620: number analyzed (Participants) | 620
  Year 2-3, n= 620 | 441
  Year 3-4,n= 514: number analyzed (Participants) | 514
  Year 3-4,n= 514 | 344
  Year 4-5,n= 442: number analyzed (Participants) | 442
  Year 4-5,n= 442 | 261
  Year 5-6, n =345: number analyzed (Participants) | 345
  Year 5-6, n =345 | 181
  Year 6-7, n= 219: number analyzed (Participants) | 219
  Year 6-7, n= 219 | 92
  Year 7-8, n = 65: number analyzed (Participants) | 65
  Year 7-8, n = 65 | 26
  Year 8 plus,n = 6: number analyzed (Participants) | 6
  Year 8 plus,n = 6 | 3

2. Primary Outcome: AE Rates by System Organ Class (SOC) During the Study
Description: AE rates by SOC adjusting for participant-years on study drug anytime post Baseline are summarized, which included the follow up visits. Only treatment-emergent AEs are summarized. The event rate of an AE was calculated as the number of events per 100 participant years. Participant years were calculated as sum across all participants ([last visit of interval day - first visit of interval day + 1] divided by365). Participant years excluded between study gaps if participant had not started extension study on date of last visit of parent study.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Adverse events per 100 participant years
Units Other Than Participants: Subject years
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Number analyzed (Subject years) | 3352
Adverse events per 100 participant years
  Infections and infestations | 101.8
  Gastrointestinal disorders | 32.8
  Musculoskeletal and connective tissuedisorder | 32.8
  Nervous system disorders | 22.6
  Skin and subcutaneous and tissue disorders | 22.5
  Respiratory,thoracic and mediastinal disorder | 14.9
  Vascular disorders | 13.3
  General disorders and administration sitecondition | 11.8
  Injury, poisoning andprocedural complications | 11.5
  Blood and lymphatic system disorders | 7.5
  Eye disorders | 6.6
  Reproductive system and breast disorders | 6.4
  Investigations | 5.8
  Psychiatric disorders | 5.6
  Renal and urinary and disorder | 5.3
  Metabolism and nutrition disorder | 3.6
  Cardiac disorders | 3.0
  Ear and labyrinth disorder | 2.4
  Neoplasms benign,malignant andunspecified | 2.2
  Hepatobiliary disorders | 1.8
  Immune system disorder | 1.2
  Endocrine disorders | 1.0
  Social circumstances | 0.7
  Congenital, familial and genetic disorders | 0.1
  Pregnancy, puerperium and perinatal conditions | 0.1
  Product Issues | 0.1

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: An adverse event resulting in death, is life threatening (ie, an immediate threat to life), inpatient hospitalization, prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or any other situation which is medically important is categorized as SAE. Only treatment-emergent AEs are summarized.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Participants
  Any post-Baseline,n=735 | 231
  Year 0-1,n=735 | 78
  Year 1-2,n = 701: number analyzed (Participants) | 701
  Year 1-2,n = 701 | 58
  Year 2-3,n = 620: number analyzed (Participants) | 620
  Year 2-3,n = 620 | 66
  Year 3-4,n= 514: number analyzed (Participants) | 514
  Year 3-4,n= 514 | 44
  Year 4-5 ,n= 442: number analyzed (Participants) | 442
  Year 4-5 ,n= 442 | 27
  Year 5-6,n=345: number analyzed (Participants) | 345
  Year 5-6,n=345 | 16
  Year 6-7,n= 219: number analyzed (Participants) | 219
  Year 6-7,n= 219 | 11
  Year 7-8,n= 65: number analyzed (Participants) | 65
  Year 7-8,n= 65 | 1
  Year 8 plus,n= 6: number analyzed (Participants) | 6
  Year 8 plus,n= 6 | 0

4. Primary Outcome: SAE Rates by SOC During the Study
Description: SAE rates by SOC adjusting for participants-years on study drug anytime post Baseline are summarized, which included the follow up visits. Only treatment-emergent SAEs are summarized. The event rate of an SAE was calculated as the number of events per 100 participant years. Participants years were calculated as = sum across all participants ([last visit of interval day - first visit of interval day + 1] divided by 365). Participants years excluded between study gaps if participant had not started extension study on date of last visit of parent study.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Adverse events per 100 participant years
Units Other Than Participants: Subject years
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Number analyzed (Subject years) | 3352
Adverse events per 100 participant years
  Infections and infestations | 5.1
  Blood and lymphatic system disorders | 1.0
  Musculoskeletal and connective tissue disorder | 1.0
  Gastrointestinal disorders | 1.0
  Renal and urinary disorders | 0.8
  Vascular disorders | 0.8
  Injury, poisoning andprocedural complications | 0.8
  General disorders and administration sitecondition | 0.6
  Nervous system disorders | 0.6
  Respiratory, thoracic and mediastinal disorder | 0.5
  Cardiac disorders | 0.5
  Skin and subcutaneous tissue disorders | 0.5
  Neoplasms benign, malignant and unspecified | 0.4
  Reproductive system and breast disorder | 0.4
  Psychiatric disorders | 0.4
  Hepatobiliary disorders | 0.3
  Metabolism and nutrition disorders | 0.1
  Pregnancy, puerperium and perinatal condition | 0.1
  Endocrine disorders | 0.1
  Immune system disorders | 0.1
  Ear and labyrinth disorders | 0.1
  Eye disorders | 0.1

5. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (APTT) and Prothrombin Time (PT) at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 hematology parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in APTT and PT is summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Seconds
  Year1,Week4,APTT,n=208: number analyzed (Participants) | 208
  Year1,Week4,APTT,n=208 | 0.7 (5.27)
  Year1,Week12,APTT,n=208: number analyzed (Participants) | 208
  Year1,Week12,APTT,n=208 | 2.1 (12.31)
  Year1,Week24,APTT,n=686: number analyzed (Participants) | 686
  Year1,Week24,APTT,n=686 | 0.1 (9.10)
  Year1,Week36,APTT,n=193: number analyzed (Participants) | 193
  Year1,Week36,APTT,n=193 | 2.5 (5.75)
  Year1,Week48,APTT,n=666: number analyzed (Participants) | 666
  Year1,Week48,APTT,n=666 | 0.8 (9.48)
  Year2,Week24,APTT,n=625: number analyzed (Participants) | 625
  Year2,Week24,APTT,n=625 | 2.7 (9.74)
  Year2,Week48,APTT,n=572: number analyzed (Participants) | 572
  Year2,Week48,APTT,n=572 | 2.7 (9.66)
  Year3,Week24,APTT,n=521: number analyzed (Participants) | 521
  Year3,Week24,APTT,n=521 | 3.4 (10.01)
  Year3,Week48,APTT,n=470: number analyzed (Participants) | 470
  Year3,Week48,APTT,n=470 | 3.9 (11.41)
  Year4,Week24,APTT,n=422: number analyzed (Participants) | 422
  Year4,Week24,APTT,n=422 | 3.5 (10.70)
  Year4,Week48,APTT,n=412: number analyzed (Participants) | 412
  Year4,Week48,APTT,n=412 | 4.2 (6.63)
  Year5,Week24,APTT,n=383: number analyzed (Participants) | 383
  Year5,Week24,APTT,n=383 | 4.1 (10.71)
  Year5,Week48,APTT,n=349: number analyzed (Participants) | 349
  Year5,Week48,APTT,n=349 | 3.5 (6.35)
  Year6,Week24,APTT,n=292: number analyzed (Participants) | 292
  Year6,Week24,APTT,n=292 | 3.8 (6.58)
  Year6,Week48,APTT,n=277: number analyzed (Participants) | 277
  Year6,Week48,APTT,n=277 | 4.3 (7.91)
  Year7,Week24,APTT,n=177: number analyzed (Participants) | 177
  Year7,Week24,APTT,n=177 | 6.4 (14.52)
  Year7,Week48,APTT,n=131: number analyzed (Participants) | 131
  Year7,Week48,APTT,n=131 | 4.1 (6.23)
  Year8,Week24,APTT,n=52: number analyzed (Participants) | 52
  Year8,Week24,APTT,n=52 | 5.6 (7.54)
  Year8,Week48,APTT,n=13: number analyzed (Participants) | 13
  Year8,Week48,APTT,n=13 | 4.2 (3.98)
  Year9,Week24,APTT,n=6: number analyzed (Participants) | 6
  Year9,Week24,APTT,n=6 | 5.0 (6.39)
  Year9,Week48,APTT,n=1: number analyzed (Participants) | 1
  Year9,Week48,APTT,n=1 | 9.0 (NA) — NA indicates standard deviation was not calculable for a single data point
  Exit, APTT,n=586: number analyzed (Participants) | 586
  Exit, APTT,n=586 | 3.2 (10.71)
  8 Week,Follow up,n=524: number analyzed (Participants) | 524
  8 Week,Follow up,n=524 | 3.4 (8.14)
  Year1,Week4,PT,n=205: number analyzed (Participants) | 205
  Year1,Week4,PT,n=205 | -0.22 (5.139)
  Year1,Week12,PT,n=206: number analyzed (Participants) | 206
  Year1,Week12,PT,n=206 | 1.71 (19.533)
  Year1,Week24,PT,n=686: number analyzed (Participants) | 686
  Year1,Week24,PT,n=686 | -0.43 (8.267)
  Year1,Week36,PT,n=193: number analyzed (Participants) | 193
  Year1,Week36,PT,n=193 | 0.13 (3.357)
  Year1,Week48,PT,n=666: number analyzed (Participants) | 666
  Year1,Week48,PT,n=666 | -0.45 (8.174)
  Year2,Week24,PT,n=626: number analyzed (Participants) | 626
  Year2,Week24,PT,n=626 | 0.15 (11.528)
  Year2,Week48,PT,n=572: number analyzed (Participants) | 572
  Year2,Week48,PT,n=572 | -0.26 (8.925)
  Year3,Week24,PT,n=521: number analyzed (Participants) | 521
  Year3,Week24,PT,n=521 | 0.12 (9.609)
  Year3,Week48,PT,n=469: number analyzed (Participants) | 469
  Year3,Week48,PT,n=469 | 0.63 (14.334)
  Year4,Week24,PT,n=422: number analyzed (Participants) | 422
  Year4,Week24,PT,n=422 | 0.06 (10.458)
  Year4,Week48,PT,n=412: number analyzed (Participants) | 412
  Year4,Week48,PT,n=412 | 0.40 (4.228)
  Year5,Week24,PT,n=384: number analyzed (Participants) | 384
  Year5,Week24,PT,n=384 | -0.14 (10.810)
  Year5,Week48,PT,n=349: number analyzed (Participants) | 349
  Year5,Week48,PT,n=349 | 0.61 (11.276)
  Year6,Week24,PT,n=292: number analyzed (Participants) | 292
  Year6,Week24,PT,n=292 | 0.64 (8.023)
  Year6,Week48,PT,n=278: number analyzed (Participants) | 278
  Year6,Week48,PT,n=278 | 0.85 (12.414)
  Year7,Week24,PT,n=177: number analyzed (Participants) | 177
  Year7,Week24,PT,n=177 | 1.76 (14.272)
  Year7,Week48,PT,n=131: number analyzed (Participants) | 131
  Year7,Week48,PT,n=131 | 0.36 (2.290)
  Year8,Week24,PT,n=52: number analyzed (Participants) | 52
  Year8,Week24,PT,n=52 | 1.21 (6.716)
  Year8,Week48,PT,n=13: number analyzed (Participants) | 13
  Year8,Week48,PT,n=13 | 0.52 (0.600)
  Year9,Week24,PT,n=6: number analyzed (Participants) | 6
  Year9,Week24,PT,n=6 | 0.50 (0.657)
  Year9,Week48,PT,n=1: number analyzed (Participants) | 1
  Year9,Week48,PT,n=1 | 1.00 (NA) — NA indicates standard deviation was not calculable for a single data point
  Exit,PT, n=587: number analyzed (Participants) | 587
  Exit,PT, n=587 | 0.25 (9.973)
  8 Week, Follow up,n=524: number analyzed (Participants) | 524
  8 Week, Follow up,n=524 | 0.50 (4.965)

6. Primary Outcome: Change From Baseline in Platelets (Plt), Lymphocytes (Lymp), Leukocytes (Leu), Eosinophils (Eos), Basophils (Baso), Monocytes (Mono), Neutrophils (Neu), Neutrophils Band Form (NeuBF), Neutrophils Segmented (NeuS) at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 hematology parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Plt, Lymp, Leu, Eos, Baso, Mono, Neu, NeuBF, and NueS are summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Billion cells per liter
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Billion cells per liter
  Baso,Year1,Week4,n=693: number analyzed (Participants) | 693
  Baso,Year1,Week4,n=693 | 0.002 (0.0172)
  Baso,Year1,Week12,n=694: number analyzed (Participants) | 694
  Baso,Year1,Week12,n=694 | 0.002 (0.0187)
  Baso,Year1,Week24,n=696: number analyzed (Participants) | 696
  Baso,Year1,Week24,n=696 | 0.002 (0.0176)
  Baso,Year1,Week36,n=682: number analyzed (Participants) | 682
  Baso,Year1,Week36,n=682 | 0.002 (0.0179)
  Baso,Year1,Week48,n=684: number analyzed (Participants) | 684
  Baso,Year1,Week48,n=684 | 0.003 (0.0183)
  Baso,Year2,Week24,n=629: number analyzed (Participants) | 629
  Baso,Year2,Week24,n=629 | 0.004 (0.0190)
  Baso,Year2,Week48,n=589: number analyzed (Participants) | 589
  Baso,Year2,Week48,n=589 | 0.004 (0.0200)
  Baso,Year3,Week24,n=533: number analyzed (Participants) | 533
  Baso,Year3,Week24,n=533 | 0.005 (0.0165)
  Baso,Year3,Week48,n=476: number analyzed (Participants) | 476
  Baso,Year3,Week48,n=476 | 0.008 (0.0194)
  Baso,Year4,Week24,n=446: number analyzed (Participants) | 446
  Baso,Year4,Week24,n=446 | 0.007 (0.0192)
  Baso,Year4,Week48,n=423: number analyzed (Participants) | 423
  Baso,Year4,Week48,n=423 | 0.008 (0.0202)
  Baso,Year5,Week24,n=389: number analyzed (Participants) | 389
  Baso,Year5,Week24,n=389 | 0.007 (0.0191)
  Baso,Year5,Week48,n=360: number analyzed (Participants) | 360
  Baso,Year5,Week48,n=360 | 0.005 (0.0191)
  Baso,Year6,Week24,n=306: number analyzed (Participants) | 306
  Baso,Year6,Week24,n=306 | 0.006 (0.0184)
  Baso,Year6,Week48,n=282: number analyzed (Participants) | 282
  Baso,Year6,Week48,n=282 | 0.007 (0.0198)
  Baso,Year7,Week24,n=181: number analyzed (Participants) | 181
  Baso,Year7,Week24,n=181 | 0.007 (0.0211)
  Baso,Year7,Week48,n=130: number analyzed (Participants) | 130
  Baso,Year7,Week48,n=130 | 0.012 (0.0259)
  Baso,Year8,Week24,n=52: number analyzed (Participants) | 52
  Baso,Year8,Week24,n=52 | 0.014 (0.0187)
  Baso,Year8,Week48,n=13: number analyzed (Participants) | 13
  Baso,Year8,Week48,n=13 | 0.001 (0.0166)
  Baso,Year9,Week24,n=6: number analyzed (Participants) | 6
  Baso,Year9,Week24,n=6 | 0.003 (0.0082)
  Baso,Year9,Week48,n=1: number analyzed (Participants) | 1
  Baso,Year9,Week48,n=1 | 0.010 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Baso,Exit,n=614: number analyzed (Participants) | 614
  Baso,Exit,n=614 | 0.005 (0.0204)
  Baso,8 Week,Follow up,n=532: number analyzed (Participants) | 532
  Baso,8 Week,Follow up,n=532 | 0.009 (0.0253)
  Eos,Year1,Week4,n=693: number analyzed (Participants) | 693
  Eos,Year1,Week4,n=693 | 0.007 (0.1597)
  Eos,Year1,Week12,n=694: number analyzed (Participants) | 694
  Eos,Year1,Week12,n=694 | 0.003 (0.1595)
  Eos,Year1,Week24,n=696: number analyzed (Participants) | 696
  Eos,Year1,Week24,n=696 | 0.000 (0.1614)
  Eos,Year1,Week36,n=682: number analyzed (Participants) | 682
  Eos,Year1,Week36,n=682 | 0.020 (0.1866)
  Eos,Year1,Week48,n=684: number analyzed (Participants) | 684
  Eos,Year1,Week48,n=684 | 0.001 (0.1763)
  Eos,Year2,Week24,n=629: number analyzed (Participants) | 629
  Eos,Year2,Week24,n=629 | 0.004 (0.1605)
  Eos,Year2,Week48,n=589: number analyzed (Participants) | 589
  Eos,Year2,Week48,n=589 | -0.004 (0.1858)
  Eos,Year3,Week24,n=533: number analyzed (Participants) | 533
  Eos,Year3,Week24,n=533 | -0.011 (0.2074)
  Eos,Year3,Week48,n=476: number analyzed (Participants) | 476
  Eos,Year3,Week48,n=476 | -0.026 (0.2053)
  Eos,Year4,Week24,n=446: number analyzed (Participants) | 446
  Eos,Year4,Week24,n=446 | -0.041 (0.1792)
  Eos,Year4,Week48,n=423: number analyzed (Participants) | 423
  Eos,Year4,Week48,n=423 | -0.047 (0.1676)
  Eos,Year5,Week24,n=389: number analyzed (Participants) | 389
  Eos,Year5,Week24,n=389 | -0.035 (0.1949)
  Eos,Year5,Week48,n=360: number analyzed (Participants) | 360
  Eos,Year5,Week48,n=360 | -0.045 (0.1807)
  Eos,Year6,Week24,n=306: number analyzed (Participants) | 306
  Eos,Year6,Week24,n=306 | -0.046 (0.1801)
  Eos,Year6,Week48,n=282: number analyzed (Participants) | 282
  Eos,Year6,Week48,n=282 | -0.037 (0.1976)
  Eos,Year7,Week24,n=181: number analyzed (Participants) | 181
  Eos,Year7,Week24,n=181 | -0.046 (0.1710)
  Eos,Year7,Week48,n=130: number analyzed (Participants) | 130
  Eos,Year7,Week48,n=130 | -0.020 (0.2276)
  Eos,Year8,Week24,n=52: number analyzed (Participants) | 52
  Eos,Year8,Week24,n=52 | -0.017 (0.1753)
  Eos,Year8,Week48,n=13: number analyzed (Participants) | 13
  Eos,Year8,Week48,n=13 | -0.041 (0.1130)
  Eos,Year9,Week24,n=6: number analyzed (Participants) | 6
  Eos,Year9,Week24,n=6 | -0.088 (0.1078)
  Eos,Year9,Week48,n=1: number analyzed (Participants) | 1
  Eos,Year9,Week48,n=1 | -0.040 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Eos, Exit, n=614: number analyzed (Participants) | 614
  Eos, Exit, n=614 | -0.026 (0.1754)
  Eso, 8 Week Follow up, n=532: number analyzed (Participants) | 532
  Eso, 8 Week Follow up, n=532 | -0.030 (0.1920)
  Leu,Year1,Week4,n=696: number analyzed (Participants) | 696
  Leu,Year1,Week4,n=696 | 0.16 (1.928)
  Leu,Year1,Week12,n=697: number analyzed (Participants) | 697
  Leu,Year1,Week12,n=697 | 0.19 (2.106)
  Leu,Year1,Week24,n=697: number analyzed (Participants) | 697
  Leu,Year1,Week24,n=697 | 0.04 (2.142)
  Leu,Year1,Week36,n=682: number analyzed (Participants) | 682
  Leu,Year1,Week36,n=682 | 0.05 (2.190)
  Leu,Year1,Week48,n=684: number analyzed (Participants) | 684
  Leu,Year1,Week48,n=684 | 0.02 (2.274)
  Leu,Year2,Week24,n=630: number analyzed (Participants) | 630
  Leu,Year2,Week24,n=630 | -0.19 (2.287)
  Leu,Year2,Week48,n=589: number analyzed (Participants) | 589
  Leu,Year2,Week48,n=589 | -0.11 (2.449)
  Leu,Year3,Week24,n=533: number analyzed (Participants) | 533
  Leu,Year3,Week24,n=533 | -0.03 (2.544)
  Leu,Year3,Week24,n=476: number analyzed (Participants) | 476
  Leu,Year3,Week24,n=476 | 0.06 (2.393)
  Leu,Year4,Week24,n=446: number analyzed (Participants) | 446
  Leu,Year4,Week24,n=446 | -0.01 (2.520)
  Leu,Year4,Week48,n=423: number analyzed (Participants) | 423
  Leu,Year4,Week48,n=423 | -0.06 (2.661)
  Leu,Year5,Week24,n=389: number analyzed (Participants) | 389
  Leu,Year5,Week24,n=389 | 0.05 (2.430)
  Leu,Year5,Week48,n=360: number analyzed (Participants) | 360
  Leu,Year5,Week48,n=360 | -0.06 (2.463)
  Leu,Year6,Week24,n=306: number analyzed (Participants) | 306
  Leu,Year6,Week24,n=306 | 0.04 (2.449)
  Leu,Year6,Week48,n=282: number analyzed (Participants) | 282
  Leu,Year6,Week48,n=282 | 0.17 (2.579)
  Leu,Year7,Week24,n=181: number analyzed (Participants) | 181
  Leu,Year7,Week24,n=181 | 0.12 (2.395)
  Leu,Year7,Week48,n=130: number analyzed (Participants) | 130
  Leu,Year7,Week48,n=130 | 0.48 (2.354)
  Leu,Year8,Week24,n=52: number analyzed (Participants) | 52
  Leu,Year8,Week24,n=52 | 0.38 (2.761)
  Leu,Year8,Week48,n=13: number analyzed (Participants) | 13
  Leu,Year8,Week48,n=13 | -0.65 (3.136)
  Leu,Year9,Week24,n=6: number analyzed (Participants) | 6
  Leu,Year9,Week24,n=6 | -0.35 (3.422)
  Leu,Year9,Week48,n=1: number analyzed (Participants) | 1
  Leu,Year9,Week48,n=1 | -3.90 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Leu, Exit, n=614: number analyzed (Participants) | 614
  Leu, Exit, n=614 | 0.18 (2.650)
  Leu, 8 Week Follow up,n=532: number analyzed (Participants) | 532
  Leu, 8 Week Follow up,n=532 | 0.21 (2.496)
  Lymp,Year1,Week4,n=693: number analyzed (Participants) | 693
  Lymp,Year1,Week4,n=693 | 0.093 (0.5986)
  Lymp,Year1,Week12,n=694: number analyzed (Participants) | 694
  Lymp,Year1,Week12,n=694 | 0.107 (0.6607)
  Lymp,Year1,Week24,n=696: number analyzed (Participants) | 696
  Lymp,Year1,Week24,n=696 | 0.066 (0.6544)
  Lymp,Year1,Week36,n=682: number analyzed (Participants) | 682
  Lymp,Year1,Week36,n=682 | 0.119 (0.6583)
  Lymp,Year1,Week48,n=684: number analyzed (Participants) | 684
  Lymp,Year1,Week48,n=684 | 0.048 (0.6361)
  Lymp,Year2,Week24,n=629: number analyzed (Participants) | 629
  Lymp,Year2,Week24,n=629 | 0.051 (0.6898)
  Lymp,Year2,Week48,n=589: number analyzed (Participants) | 589
  Lymp,Year2,Week48,n=589 | 0.067 (0.6971)
  Lymp,Year3,Week24,n=533: number analyzed (Participants) | 533
  Lymp,Year3,Week24,n=533 | 0.057 (0.6717)
  Lymp,Year3,Week48,n=476: number analyzed (Participants) | 476
  Lymp,Year3,Week48,n=476 | 0.038 (0.6676)
  Lymp,Year4,Week24,n=446: number analyzed (Participants) | 446
  Lymp,Year4,Week24,n=446 | 0.054 (0.6858)
  Lymp,Year4,Week48,n=423: number analyzed (Participants) | 423
  Lymp,Year4,Week48,n=423 | 0.067 (0.7186)
  Lymp,Year5,Week24,n=389: number analyzed (Participants) | 389
  Lymp,Year5,Week24,n=389 | 0.023 (0.6810)
  Lymp,Year5,Week48,n=360: number analyzed (Participants) | 360
  Lymp,Year5,Week48,n=360 | 0.078 (0.7485)
  Lymp,Year6,Week24,n=306: number analyzed (Participants) | 306
  Lymp,Year6,Week24,n=306 | 0.147 (0.7251)
  Lymp,Year6,Week48,n=282: number analyzed (Participants) | 282
  Lymp,Year6,Week48,n=282 | 0.168 (0.7523)
  Lymp,Year7,Week24,n=181: number analyzed (Participants) | 181
  Lymp,Year7,Week24,n=181 | 0.175 (0.7670)
  Lymp,Year7,Week48,n=130: number analyzed (Participants) | 130
  Lymp,Year7,Week48,n=130 | 0.169 (0.6639)
  Lymp,Year8,Week24,n=52: number analyzed (Participants) | 52
  Lymp,Year8,Week24,n=52 | 0.300 (0.7553)
  Lymp,Year8,Week48,n=13: number analyzed (Participants) | 13
  Lymp,Year8,Week48,n=13 | 0.052 (0.5252)
  Lymp,Year9,Week24,n=6: number analyzed (Participants) | 6
  Lymp,Year9,Week24,n=6 | -0.032 (0.6156)
  Lymp,Year9,Week48,n=1: number analyzed (Participants) | 1
  Lymp,Year9,Week48,n=1 | -0.460 (NA) — NA indicates standard deviation was not calculable for a single data point
  Lymp,Exit,n=614: number analyzed (Participants) | 614
  Lymp,Exit,n=614 | 0.128 (0.7808)
  Lymp,8 Week Follow up,n=532: number analyzed (Participants) | 532
  Lymp,8 Week Follow up,n=532 | 0.140 (0.7453)
  Mono,Year1,Week4,n=693: number analyzed (Participants) | 693
  Mono,Year1,Week4,n=693 | 0.025 (0.2108)
  Mono,Year1,Week12,n=694: number analyzed (Participants) | 694
  Mono,Year1,Week12,n=694 | 0.036 (0.2043)
  Mono,Year1,Week24,n=696: number analyzed (Participants) | 696
  Mono,Year1,Week24,n=696 | 0.028 (0.2127)
  Mono,Year1,Week36,n=682: number analyzed (Participants) | 682
  Mono,Year1,Week36,n=682 | 0.053 (0.2053)
  Mono,Year1,Week48,n=684: number analyzed (Participants) | 684
  Mono,Year1,Week48,n=684 | 0.050 (0.2069)
  Mono,Year2,Week24,n=629: number analyzed (Participants) | 629
  Mono,Year2,Week24,n=629 | 0.034 (0.1992)
  Mono,Year2,Week48,n=589: number analyzed (Participants) | 589
  Mono,Year2,Week48,n=589 | 0.050 (0.2172)
  Mono,Year3,Week24,n=533: number analyzed (Participants) | 533
  Mono,Year3,Week24,n=533 | 0.053 (0.2314)
  Mono,Year3,Week48,n=476: number analyzed (Participants) | 476
  Mono,Year3,Week48,n=476 | 0.084 (0.1994)
  Mono,Year4,Week24,n=446: number analyzed (Participants) | 446
  Mono,Year4,Week24,n=446 | 0.071 (0.2085)
  Mono,Year4,Week48,n=423: number analyzed (Participants) | 423
  Mono,Year4,Week48,n=423 | 0.076 (0.2040)
  Mono,Year5,Week24,n=389: number analyzed (Participants) | 389
  Mono,Year5,Week24,n=389 | 0.089 (0.2015)
  Mono,Year5,Week48,n=360: number analyzed (Participants) | 360
  Mono,Year5,Week48,n=360 | 0.088 (0.2044)
  Mono,Year6,Week24,n=306: number analyzed (Participants) | 306
  Mono,Year6,Week24,n=306 | 0.087 (0.2043)
  Mono,Year6,Week48,n=282: number analyzed (Participants) | 282
  Mono,Year6,Week48,n=282 | 0.086 (0.2063)
  Mono,Year7,Week24,n=181: number analyzed (Participants) | 181
  Mono,Year7,Week24,n=181 | 0.113 (0.2155)
  Mono,Year7,Week48,n=130: number analyzed (Participants) | 130
  Mono,Year7,Week48,n=130 | 0.134 (0.2090)
  Mono,Year8,Week24,n=52: number analyzed (Participants) | 52
  Mono,Year8,Week24,n=52 | 0.173 (0.2014)
  Mono,Year8,Week48,n=13: number analyzed (Participants) | 13
  Mono,Year8,Week48,n=13 | 0.021 (0.1503)
  Mono,Year9,Week24,n=6: number analyzed (Participants) | 6
  Mono,Year9,Week24,n=6 | 0.022 (0.1931)
  Mono,Year9,Week48,n=1: number analyzed (Participants) | 1
  Mono,Year9,Week48,n=1 | -0.120 (NA) — NA indicates standard deviation was not calculable for a single data point
  Mono, Exit,n=614: number analyzed (Participants) | 614
  Mono, Exit,n=614 | 0.083 (0.2157)
  Mono, 8 Week Follow up, n=532: number analyzed (Participants) | 532
  Mono, 8 Week Follow up, n=532 | 0.084 (0.2189)
  Neu,Yaer1,Week4,n=688: number analyzed (Participants) | 688
  Neu,Yaer1,Week4,n=688 | 0.024 (2.0482)
  Neru,Year1,Week12,n=690: number analyzed (Participants) | 690
  Neru,Year1,Week12,n=690 | 0.047 (2.1575)
  Neu,Year1,Week24,n=691: number analyzed (Participants) | 691
  Neu,Year1,Week24,n=691 | -0.059 (2.1845)
  Neu,Year1,Week36,n=677: number analyzed (Participants) | 677
  Neu,Year1,Week36,n=677 | -0.141 (2.1907)
  Neu,Year1,Week48,n=679: number analyzed (Participants) | 679
  Neu,Year1,Week48,n=679 | -0.078 (2.3164)
  Neu,Year2,Week24,n=624: number analyzed (Participants) | 624
  Neu,Year2,Week24,n=624 | -0.286 (2.2746)
  Neu,Year2,Week48,n=584: number analyzed (Participants) | 584
  Neu,Year2,Week48,n=584 | -0.230 (2.3963)
  Neu,Year3,Week24,n=528: number analyzed (Participants) | 528
  Neu,Year3,Week24,n=528 | -0.135 (2.4914)
  Neu,Year3,Week48,n=471: number analyzed (Participants) | 471
  Neu,Year3,Week48,n=471 | -0.049 (2.3683)
  Neu,Year4,Week24,n=446: number analyzed (Participants) | 446
  Neu,Year4,Week24,n=446 | -0.104 (2.3846)
  Neu,Year4,Week48,n=423: number analyzed (Participants) | 423
  Neu,Year4,Week48,n=423 | -0.160 (2.5563)
  Neu,Year5,Week24,n=384: number analyzed (Participants) | 384
  Neu,Year5,Week24,n=384 | -0.031 (2.3060)
  Neu,Year5,Week48,n=356: number analyzed (Participants) | 356
  Neu,Year5,Week48,n=356 | -0.198 (2.3952)
  Neu,Year6,Week24,n=306: number analyzed (Participants) | 306
  Neu,Year6,Week24,n=306 | -0.151 (2.3083)
  Neu,Year6,Week48,n=282: number analyzed (Participants) | 282
  Neu,Year6,Week48,n=282 | -0.060 (2.4314)
  Neu,Year7,Week24,n=181: number analyzed (Participants) | 181
  Neu,Year7,Week24,n=181 | -0.129 (2.3908)
  Neu,Year7,Week48,n=130: number analyzed (Participants) | 130
  Neu,Year7,Week48,n=130 | -0.687 (3.0412)
  Neu,Year8,Week24,n=52: number analyzed (Participants) | 52
  Neu,Year8,Week24,n=52 | -0.092 (2.3908)
  Neu,Year8,Week48,n=13: number analyzed (Participants) | 13
  Neu,Year8,Week48,n=13 | -0.687 (3.0412)
  Neu,Year9,Week24,n=6: number analyzed (Participants) | 6
  Neu,Year9,Week24,n=6 | -0.257 (2.9192)
  Neu,Year9,Week48,n=1 | -3.300 (NA) — NA indicates standard deviation was not calculable for a single data point
  Neu, Exit, n=609: number analyzed (Participants) | 609
  Neu, Exit, n=609 | -0.006 (2.5612)
  Neu,8 Week Follow up,n=528: number analyzed (Participants) | 528
  Neu,8 Week Follow up,n=528 | 0.001 (2.3935)
  NeuBF,Year1,Week4,n=4: number analyzed (Participants) | 4
  NeuBF,Year1,Week4,n=4 | 0.013 (0.1473)
  NeuBF,Year1,Week12,n=4: number analyzed (Participants) | 4
  NeuBF,Year1,Week12,n=4 | 0.073 (0.1106)
  NeuBF,Year1,Week24,n=5: number analyzed (Participants) | 5
  NeuBF,Year1,Week24,n=5 | -0.000 (0.2699)
  NeuBF,Year1,Week36,n=4: number analyzed (Participants) | 4
  NeuBF,Year1,Week36,n=4 | 0.045 (0.0465)
  NeuBF,Year1,Week48,n=2: number analyzed (Participants) | 2
  NeuBF,Year1,Week48,n=2 | 0.105 (0.1909)
  NeuBF,Year2,Week24,n=1: number analyzed (Participants) | 1
  NeuBF,Year2,Week24,n=1 | 0.120 (NA) — NA indicates standard deviation was not calculable for a single data point.
  NeuBF,Year2,Week48,n=0: number analyzed (Participants) | 0
  NeuBF,Year3,Week24,n=1: number analyzed (Participants) | 1
  NeuBF,Year3,Week24,n=1 | 0.070 (NA) — NA indicates standard deviation was not calculable for a single data point.
  NeuBF,Year3,Week48,n=0: number analyzed (Participants) | 0
  NeuBF,Year7,Week24,n=0: number analyzed (Participants) | 0
  NeuBF,Exit,n=2: number analyzed (Participants) | 2
  NeuBF,Exit,n=2 | 0.465 (0.6435)
  NeuS,Year1,Week4,n=693: number analyzed (Participants) | 693
  NeuS,Year1,Week4,n=693 | 0.021 (2.0450)
  NeuS,Year1,Week12,n=694: number analyzed (Participants) | 694
  NeuS,Year1,Week12,n=694 | 0.051 (2.1519)
  NeuS,Year1,Week24,n=696: number analyzed (Participants) | 696
  NeuS,Year1,Week24,n=696 | -0.055 (2.1757)
  NeuS,Year1,Week36,n=682: number analyzed (Participants) | 682
  NeuS,Year1,Week36,n=682 | -0.139 (2.1819)
  NeuS,Year1,Week48,n=684: number analyzed (Participants) | 684
  NeuS,Year1,Week48,n=684 | -0.079 (2.3128)
  NeuS,Year2,Week24,n=629: number analyzed (Participants) | 629
  NeuS,Year2,Week24,n=629 | -0.289 (2.2609)
  NeuS,Year2,Week48,n=589: number analyzed (Participants) | 589
  NeuS,Year2,Week48,n=589 | -0.226 (2.3846)
  NeuS,Year3,Week24,n=533: number analyzed (Participants) | 533
  NeuS,Year3,Week24,n=533 | -0.130 (2.4736)
  NeuS,Year3,Week48,n=476: number analyzed (Participants) | 476
  NeuS,Year3,Week48,n=476 | -0.041 (2.3547)
  NeuS,Year4,Week24,n=446: number analyzed (Participants) | 446
  NeuS,Year4,Week24,n=446 | -0.097 (2.3804)
  NeuS,Year4,Week48,n=423: number analyzed (Participants) | 423
  NeuS,Year4,Week48,n=423 | -0.158 (2.5542)
  NeuS,Year5,Week24,n=389: number analyzed (Participants) | 389
  NeuS,Year5,Week24,n=389 | -0.024 (2.2893)
  NeuS,Year5,Week48,n=360: number analyzed (Participants) | 360
  NeuS,Year5,Week48,n=360 | -0.184 (2.3831)
  NeuS,Year6,Week24,n=306: number analyzed (Participants) | 306
  NeuS,Year6,Week24,n=306 | -0.147 (2.3029)
  NeuS,Year6,Week48,n=282: number analyzed (Participants) | 282
  NeuS,Year6,Week48,n=282 | -0.058 (2.4310)
  NeuS,Year7,Week24,n=181: number analyzed (Participants) | 181
  NeuS,Year7,Week24,n=181 | -0.151 (2.2248)
  NeuS,Year7,Week48,n=130: number analyzed (Participants) | 130
  NeuS,Year7,Week48,n=130 | 0.191 (2.2514)
  NeuS,Year8,Week24,n=52: number analyzed (Participants) | 52
  NeuS,Year8,Week24,n=52 | -0.092 (2.3908)
  NeuS,Year8,Week48,n=13: number analyzed (Participants) | 13
  NeuS,Year8,Week48,n=13 | -0.687 (3.0412)
  NeuS,Year9,Week24,n=6: number analyzed (Participants) | 6
  NeuS,Year9,Week24,n=6 | -0.257 (2.9192)
  NeuS,Year9,Week48,n=1: number analyzed (Participants) | 1
  NeuS,Year9,Week48,n=1 | -3.300 (NA) — NA indicates standard deviation was not calculable for a single data point
  NeuS,Exit,n=614: number analyzed (Participants) | 614
  NeuS,Exit,n=614 | -0.008 (2.5501)
  NeuS,8 Week Followup,n=532: number analyzed (Participants) | 532
  NeuS,8 Week Followup,n=532 | 0.007 (2.3824)
  Plt,Year1,Week4,n=683: number analyzed (Participants) | 683
  Plt,Year1,Week4,n=683 | 8.1 (38.82)
  Plt,Year1,Week12,n=690: number analyzed (Participants) | 690
  Plt,Year1,Week12,n=690 | 4.6 (43.63)
  Plt,Year1,Week24,n=687: number analyzed (Participants) | 687
  Plt,Year1,Week24,n=687 | -0.5 (47.73)
  Plt,Year1,Week36,n=680: number analyzed (Participants) | 680
  Plt,Year1,Week36,n=680 | -2.9 (50.25)
  Plt,Year1,Week48,n=677: number analyzed (Participants) | 677
  Plt,Year1,Week48,n=677 | -9.3 (50.81)
  Plt,Year2,Week24,n=631: number analyzed (Participants) | 631
  Plt,Year2,Week24,n=631 | -15.4 (53.80)
  Plt,Year2,Week48,n=583: number analyzed (Participants) | 583
  Plt,Year2,Week48,n=583 | -20.3 (56.39)
  Plt,Year3,Week24,n=526: number analyzed (Participants) | 526
  Plt,Year3,Week24,n=526 | -19.9 (57.88)
  Plt,Year3,Week48,n=476: number analyzed (Participants) | 476
  Plt,Year3,Week48,n=476 | -13.4 (65.16)
  Plt,Year4,Week24,n=441: number analyzed (Participants) | 441
  Plt,Year4,Week24,n=441 | -14.0 (59.05)
  Plt,Year4,Week48,n=420: number analyzed (Participants) | 420
  Plt,Year4,Week48,n=420 | -18.2 (63.80)
  Plt,Year5,Week24,n=388: number analyzed (Participants) | 388
  Plt,Year5,Week24,n=388 | -19.3 (61.49)
  Plt,Year5,Week48,n=360: number analyzed (Participants) | 360
  Plt,Year5,Week48,n=360 | -17.9 (63.36)
  Plt,Year6,Week24,n=305: number analyzed (Participants) | 305
  Plt,Year6,Week24,n=305 | -13.3 (61.54)
  Plt,Year6,Week48,n=282: number analyzed (Participants) | 282
  Plt,Year6,Week48,n=282 | -13.4 (60.89)
  Plt,Year7,Week24,n=181: number analyzed (Participants) | 181
  Plt,Year7,Week24,n=181 | -15.3 (63.95)
  Plt,Year7,Week48,n=130: number analyzed (Participants) | 130
  Plt,Year7,Week48,n=130 | -16.3 (70.75)
  Plt,Year8,Week24,n=52: number analyzed (Participants) | 52
  Plt,Year8,Week24,n=52 | -2.3 (80.69)
  Plt,Year8,Week48,n=13: number analyzed (Participants) | 13
  Plt,Year8,Week48,n=13 | -29.9 (88.66)
  Plt,Year9,Week24,n=6: number analyzed (Participants) | 6
  Plt,Year9,Week24,n=6 | -5.0 (82.67)
  Plt,Year9,Week48,n=1: number analyzed (Participants) | 1
  Plt,Year9,Week48,n=1 | 57.0 (NA) — NA indicates standard deviation was not calculable for a single data point
  Plt,Exit,n=613: number analyzed (Participants) | 613
  Plt,Exit,n=613 | -11.0 (64.36)
  Plt,8Week Followup,n=530: number analyzed (Participants) | 530
  Plt,8Week Followup,n=530 | -11.2 (60.57)

7. Primary Outcome: Change From Baseline in Hemoglobin (Hg) at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 hematology parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Hg is summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Gram per liter (g/L)
  Hg,Year1, Week 4,n=697: number analyzed (Participants) | 697
  Hg,Year1, Week 4,n=697 | -0.3 (7.05)
  Hg,Year1,Week12,n=698: number analyzed (Participants) | 698
  Hg,Year1,Week12,n=698 | 0.1 (8.75)
  Hg,Year1,Week24,n=699: number analyzed (Participants) | 699
  Hg,Year1,Week24,n=699 | 0.1 (9.48)
  Hg,Year1,Week36,n=688: number analyzed (Participants) | 688
  Hg,Year1,Week36,n=688 | 0.3 (9.90)
  Hg,Year1,Week48,n=686: number analyzed (Participants) | 686
  Hg,Year1,Week48,n=686 | 1.0 (11.03)
  Hg,Year2,Week24,n=635: number analyzed (Participants) | 635
  Hg,Year2,Week24,n=635 | 1.0 (11.31)
  Hg,Year2,Week48,n=591: number analyzed (Participants) | 591
  Hg,Year2,Week48,n=591 | 1.3 (12.12)
  Hg,Year3,Week24,n=534: number analyzed (Participants) | 534
  Hg,Year3,Week24,n=534 | 2.2 (12.79)
  Hg,Year3,Week48,n=478: number analyzed (Participants) | 478
  Hg,Year3,Week48,n=478 | 2.9 (12.67)
  Hg,Year4,Week24,n=446: number analyzed (Participants) | 446
  Hg,Year4,Week24,n=446 | 2.6 (12.93)
  Hg,Year,Week48,n=424: number analyzed (Participants) | 424
  Hg,Year,Week48,n=424 | 2.4 (13.59)
  Hg,Year5,Week24,n=390: number analyzed (Participants) | 390
  Hg,Year5,Week24,n=390 | 2.9 (12.76)
  Hg,Year5,Week48,n=362: number analyzed (Participants) | 362
  Hg,Year5,Week48,n=362 | 3.2 (13.26)
  Hg,Year6,Week24,n=306: number analyzed (Participants) | 306
  Hg,Year6,Week24,n=306 | 2.7 (13.19)
  Hg,Year6,Week48,n=282: number analyzed (Participants) | 282
  Hg,Year6,Week48,n=282 | 2.3 (13.83)
  Hg,Year7,Week24,n=181: number analyzed (Participants) | 181
  Hg,Year7,Week24,n=181 | 2.9 (14.54)
  Hg,Year7,Week48,n=130: number analyzed (Participants) | 130
  Hg,Year7,Week48,n=130 | 4.0 (14.66)
  Hg,Year8,Week24,n=52: number analyzed (Participants) | 52
  Hg,Year8,Week24,n=52 | 1.5 (14.84)
  Hg,Year8,Week48,n=13: number analyzed (Participants) | 13
  Hg,Year8,Week48,n=13 | -0.2 (13.95)
  Hg,Year9,Week24,n=6: number analyzed (Participants) | 6
  Hg,Year9,Week24,n=6 | -0.7 (20.67)
  Hg,Year9,Week48,n=1: number analyzed (Participants) | 1
  Hg,Year9,Week48,n=1 | -29.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Hg,Exit,n=619: number analyzed (Participants) | 619
  Hg,Exit,n=619 | 3.2 (13.90)
  Hg,8 Week Follow up,n=534: number analyzed (Participants) | 534
  Hg,8 Week Follow up,n=534 | 2.8 (13.71)

8. Primary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 hematology parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks). Change from Baseline in Hematocrit is summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Percentage of blood by volume
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Percentage of blood by volume
  Hematocrit,Year1,Week4,n=697: number analyzed (Participants) | 697
  Hematocrit,Year1,Week4,n=697 | 0.01 (2.250)
  Hematocrit,Year1,Week12,n=698: number analyzed (Participants) | 698
  Hematocrit,Year1,Week12,n=698 | 0.38 (2.729)
  Hematocrit,Year1,Week24,n=699: number analyzed (Participants) | 699
  Hematocrit,Year1,Week24,n=699 | 0.75 (2.928)
  Hematocrit,Year1,Week36,n=688: number analyzed (Participants) | 688
  Hematocrit,Year1,Week36,n=688 | 0.53 (2.954)
  Hematocrit,Year1,Week48,n=686: number analyzed (Participants) | 686
  Hematocrit,Year1,Week48,n=686 | 0.35 (3.286)
  Hematocrit,Year2,Week24,n=635: number analyzed (Participants) | 635
  Hematocrit,Year2,Week24,n=635 | 0.94 (3.427)
  Hematocrit,Year2,Week48,n=591: number analyzed (Participants) | 591
  Hematocrit,Year2,Week48,n=591 | 0.78 (3.584)
  Hematocrit,Year3,Week24,n=534: number analyzed (Participants) | 534
  Hematocrit,Year3,Week24,n=534 | 1.29 (3.828)
  Hematocrit,Year3,Week48,n=478: number analyzed (Participants) | 478
  Hematocrit,Year3,Week48,n=478 | 1.39 (3.800)
  Hematocrit,Year4,Week24,n=446: number analyzed (Participants) | 446
  Hematocrit,Year4,Week24,n=446 | 1.67 (3.834)
  Hematocrit,Year4,Week48,n=424: number analyzed (Participants) | 424
  Hematocrit,Year4,Week48,n=424 | 1.15 (3.998)
  Hematocrit,Year5,Week24,n=390: number analyzed (Participants) | 390
  Hematocrit,Year5,Week24,n=390 | 1.69 (3.776)
  Hematocrit,Year5,Week48,n=362: number analyzed (Participants) | 362
  Hematocrit,Year5,Week48,n=362 | 1.98 (3.842)
  Hematocrit,Year6,Week24,n=306: number analyzed (Participants) | 306
  Hematocrit,Year6,Week24,n=306 | 1.93 (3.939)
  Hematocrit,Year6,Week48,n=282: number analyzed (Participants) | 282
  Hematocrit,Year6,Week48,n=282 | 2.07 (4.023)
  Hematocrit,Year7,Week24,n=181: number analyzed (Participants) | 181
  Hematocrit,Year7,Week24,n=181 | 1.81 (4.251)
  Hematocrit,Year7,Week48,n=130: number analyzed (Participants) | 130
  Hematocrit,Year7,Week48,n=130 | 2.11 (4.238)
  Hematocrit,Year8,Week24,n=52: number analyzed (Participants) | 52
  Hematocrit,Year8,Week24,n=52 | 1.42 (4.390)
  Hematocrit,Year8,Week48,n=13: number analyzed (Participants) | 13
  Hematocrit,Year8,Week48,n=13 | 1.48 (4.234)
  Hematocrit,Year9,Week24,n=6: number analyzed (Participants) | 6
  Hematocrit,Year9,Week24,n=6 | 2.03 (6.001)
  Hematocrit,Year9,Week48,n=1: number analyzed (Participants) | 1
  Hematocrit,Year9,Week48,n=1 | -6.00 (NA) — NA indicates standard deviation was not calculable for a single data point
  Hematocrit,Exit,n=619: number analyzed (Participants) | 619
  Hematocrit,Exit,n=619 | 1.91 (4.202)
  Hematocrit,8 Week Follow up,n=534: number analyzed (Participants) | 534
  Hematocrit,8 Week Follow up,n=534 | 1.85 (4.077)

9. Primary Outcome: Change From Baseline in Erythrocytes (Eryth) at the Indicated Time Points
Description: Hematology parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 hematology parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Erythrocytes is summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Trillions cells per liter
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Trillions cells per liter
  Eryth,Year1,Week4,n=697: number analyzed (Participants) | 697
  Eryth,Year1,Week4,n=697 | -0.00 (0.231)
  Eryth,Year1,Week12,n=698: number analyzed (Participants) | 698
  Eryth,Year1,Week12,n=698 | 0.04 (0.280)
  Eryth,Year1,Week24,n=699: number analyzed (Participants) | 699
  Eryth,Year1,Week24,n=699 | 0.06 (0.293)
  Eryth,Year1,Week36,n=688: number analyzed (Participants) | 688
  Eryth,Year1,Week36,n=688 | 0.06 (0.299)
  Eryth,Year1,Week48,n=686: number analyzed (Participants) | 686
  Eryth,Year1,Week48,n=686 | 0.06 (0.328)
  Eryth,Year2,Week24,n=635: number analyzed (Participants) | 635
  Eryth,Year2,Week24,n=635 | 0.07 (0.335)
  Eryth,Year2,Week48,n=591: number analyzed (Participants) | 591
  Eryth,Year2,Week48,n=591 | 0.04 (0.362)
  Eryth,Year3,Week24,n=534: number analyzed (Participants) | 534
  Eryth,Year3,Week24,n=534 | 0.04 (0.364)
  Eryth,Year3,Week48,n=478: number analyzed (Participants) | 478
  Eryth,Year3,Week48,n=478 | 0.05 (0.381)
  Eryth,Year4,Week24,n=446: number analyzed (Participants) | 446
  Eryth,Year4,Week24,n=446 | 0.06 (0.372)
  Eryth,Year,Week48,n=424: number analyzed (Participants) | 424
  Eryth,Year,Week48,n=424 | 0.05 (0.379)
  Eryth,Year5,Week24,n=390: number analyzed (Participants) | 390
  Eryth,Year5,Week24,n=390 | 0.09 (0.375)
  Eryth,Year5,Week48,n=362: number analyzed (Participants) | 362
  Eryth,Year5,Week48,n=362 | 0.11 (0.383)
  Eryth,Year6,Week24,n=306: number analyzed (Participants) | 306
  Eryth,Year6,Week24,n=306 | 0.12 (0.396)
  Eryth,Year6,Week48,n=282: number analyzed (Participants) | 282
  Eryth,Year6,Week48,n=282 | 0.17 (0.408)
  Eryth,Year7,Week24,n=181: number analyzed (Participants) | 181
  Eryth,Year7,Week24,n=181 | 0.17 (0.415)
  Eryth,Year7,Week48,n=130: number analyzed (Participants) | 130
  Eryth,Year7,Week48,n=130 | 0.22 (0.387)
  Eryth,Year8,Week24,n=52: number analyzed (Participants) | 52
  Eryth,Year8,Week24,n=52 | 0.21 (0.375)
  Eryth,Year8,Week48,n=13: number analyzed (Participants) | 13
  Eryth,Year8,Week48,n=13 | 0.15 (0.207)
  Eryth,Year9,Week24,n=6: number analyzed (Participants) | 6
  Eryth,Year9,Week24,n=6 | 0.30 (0.374)
  Eryth,Year9,Week48,n=1: number analyzed (Participants) | 1
  Eryth,Year9,Week48,n=1 | 0.20 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Eryth,Exit,n=619: number analyzed (Participants) | 619
  Eryth,Exit,n=619 | 0.14 (0.431)
  Eryth,8 Week Follow up,n=534: number analyzed (Participants) | 534
  Eryth,8 Week Follow up,n=534 | 0.13 (0.411)

10. Primary Outcome: Change From Baseline in Calcium (Ca), Carbon Dioxide (CO2), Chloride, Magnesium (Mg), Phosphate (Phos), Potassium (K), Sodium (Na) at the Indicated Time Points
Description: Electrolytes parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 electrolytes parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Ca,CO2, Chloride, Mg, Phos, K and Na were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Millimoles per liter (mmol/L)
  Ca,Year1,Week4,n=697: number analyzed (Participants) | 697
  Ca,Year1,Week4,n=697 | 0.0030 (0.0763)
  Ca,Year1,Week12,n=696: number analyzed (Participants) | 696
  Ca,Year1,Week12,n=696 | 0.0020 (0.0749)
  Ca,Year1,Week24,n=696: number analyzed (Participants) | 696
  Ca,Year1,Week24,n=696 | -0.0035 (0.0750)
  Ca,Year1,Week36,n=677: number analyzed (Participants) | 677
  Ca,Year1,Week36,n=677 | 0.0024 (0.0836)
  Ca,Year1,Week48,n=687: number analyzed (Participants) | 687
  Ca,Year1,Week48,n=687 | -0.0065 (0.0778)
  Ca,Year2,Week24,n=636: number analyzed (Participants) | 636
  Ca,Year2,Week24,n=636 | -0.0075 (0.0764)
  Ca,Year2,Week48,n=587: number analyzed (Participants) | 587
  Ca,Year2,Week48,n=587 | -0.0091 (0.0837)
  Ca,Year3,Week24,n=526: number analyzed (Participants) | 526
  Ca,Year3,Week24,n=526 | -0.0047 (0.0810)
  Ca,Year3,Week48,n=481: number analyzed (Participants) | 481
  Ca,Year3,Week48,n=481 | -0.0123 (0.0800)
  Ca,Year4,Week24,n=438: number analyzed (Participants) | 438
  Ca,Year4,Week24,n=438 | -0.0056 (0.0771)
  Ca,Year,Week48,n=418: number analyzed (Participants) | 418
  Ca,Year,Week48,n=418 | -0.0193 (0.0805)
  Ca,Year5,Week24,n=387: number analyzed (Participants) | 387
  Ca,Year5,Week24,n=387 | -0.0129 (0.0885)
  Ca,Year5,Week48,n=358: number analyzed (Participants) | 358
  Ca,Year5,Week48,n=358 | -0.0140 (0.0919)
  Ca,Year6,Week24,n=303: number analyzed (Participants) | 303
  Ca,Year6,Week24,n=303 | -0.0053 (0.0903)
  Ca,Year6,Week48,n=283: number analyzed (Participants) | 283
  Ca,Year6,Week48,n=283 | -0.0146 (0.0870)
  Ca,Year7,Week24,n=182: number analyzed (Participants) | 182
  Ca,Year7,Week24,n=182 | -0.0076 (0.0839)
  Ca,Year7,Week48,n=130: number analyzed (Participants) | 130
  Ca,Year7,Week48,n=130 | -0.0079 (0.1172)
  Ca,Year8,Week24,n=51: number analyzed (Participants) | 51
  Ca,Year8,Week24,n=51 | 0.0003 (0.0806)
  Ca,Year8,Week48,n=13: number analyzed (Participants) | 13
  Ca,Year8,Week48,n=13 | -0.0395 (0.0611)
  Ca,Year9,Week24,n=6: number analyzed (Participants) | 6
  Ca,Year9,Week24,n=6 | -0.0402 (0.0336)
  Ca,Year9,Week48,n=1: number analyzed (Participants) | 1
  Ca,Year9,Week48,n=1 | -0.0642 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Ca,Exit,n=619: number analyzed (Participants) | 619
  Ca,Exit,n=619 | 0.0006 (0.0864)
  Ca,8 Week Follow up,n=534: number analyzed (Participants) | 534
  Ca,8 Week Follow up,n=534 | -0.0014 (0.0909)
  CO2,Year1,Week4,n=701: number analyzed (Participants) | 701
  CO2,Year1,Week4,n=701 | -0.0 (2.77)
  CO2,Year1,Week12,n=700: number analyzed (Participants) | 700
  CO2,Year1,Week12,n=700 | -0.1 (2.76)
  CO2,Year1,Week24,n=701: number analyzed (Participants) | 701
  CO2,Year1,Week24,n=701 | -0.1 (2.73)
  CO2,Year1,Week36,n=682: number analyzed (Participants) | 682
  CO2,Year1,Week36,n=682 | 0.1 (2.73)
  CO2,Year1,Week48,n=692: number analyzed (Participants) | 692
  CO2,Year1,Week48,n=692 | -0.1 (2.78)
  CO2,Year2,Week24,n=641: number analyzed (Participants) | 641
  CO2,Year2,Week24,n=641 | -0.3 (2.94)
  CO2,Year2,Week48,n=692: number analyzed (Participants) | 692
  CO2,Year2,Week48,n=692 | -0.3 (2.87)
  CO2,Year3,Week24,n=531: number analyzed (Participants) | 531
  CO2,Year3,Week24,n=531 | -0.2 (2.90)
  CO2,Year3,Week48,n=486: number analyzed (Participants) | 486
  CO2,Year3,Week48,n=486 | -0.4 (2.75)
  CO2,Year4,Week24,n=438: number analyzed (Participants) | 438
  CO2,Year4,Week24,n=438 | -0.0 (2.76)
  CO2,Year4,Week48,n=418: number analyzed (Participants) | 418
  CO2,Year4,Week48,n=418 | -0.5 (3.04)
  CO2,Year5,Week24,n=393: number analyzed (Participants) | 393
  CO2,Year5,Week24,n=393 | -0.2 (2.90)
  CO2,Year5,Week48,n=361: number analyzed (Participants) | 361
  CO2,Year5,Week48,n=361 | -0.8 (2.82)
  CO2,Year6,Week24,n=303: number analyzed (Participants) | 303
  CO2,Year6,Week24,n=303 | -0.0 (2.86)
  CO2,Year6,Week48,n=284: number analyzed (Participants) | 284
  CO2,Year6,Week48,n=284 | -0.5 (2.76)
  CO2,Year7,Week24,n=182: number analyzed (Participants) | 182
  CO2,Year7,Week24,n=182 | 0.2 (2.78)
  CO2,Year7,Week48,n=130: number analyzed (Participants) | 130
  CO2,Year7,Week48,n=130 | 0.2 (2.67)
  CO2,Year8,Week24,n=52: number analyzed (Participants) | 52
  CO2,Year8,Week24,n=52 | 1.0 (2.78)
  CO2,Year8,Week48,n=13: number analyzed (Participants) | 13
  CO2,Year8,Week48,n=13 | 0.4 (3.38)
  CO2,Year9,Week24,n=6: number analyzed (Participants) | 6
  CO2,Year9,Week24,n=6 | -0.3 (0.82)
  CO2,Year9,Week48,n=1: number analyzed (Participants) | 1
  CO2,Year9,Week48,n=1 | -3.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  CO2,Exit,n=625: number analyzed (Participants) | 625
  CO2,Exit,n=625 | -0.3 (3.00)
  CO2,8 week Follow up,n=538: number analyzed (Participants) | 538
  CO2,8 week Follow up,n=538 | -0.2 (3.00)
  Chloride,Year1,Week4,n=707: number analyzed (Participants) | 707
  Chloride,Year1,Week4,n=707 | 0.3 (2.33)
  Chloride,Year1,Week12,n=704: number analyzed (Participants) | 704
  Chloride,Year1,Week12,n=704 | 0.6 (2.56)
  Chloride,Year1,Week24,n=703: number analyzed (Participants) | 703
  Chloride,Year1,Week24,n=703 | 0.6 (2.42)
  Chloride,Year1,Week36,n=684: number analyzed (Participants) | 684
  Chloride,Year1,Week36,n=684 | 0.6 (2.47)
  Chloride,Year1,Week48,n=693: number analyzed (Participants) | 693
  Chloride,Year1,Week48,n=693 | 0.4 (2.44)
  Chloride,Year2,Week24,n=643: number analyzed (Participants) | 643
  Chloride,Year2,Week24,n=643 | 0.5 (2.62)
  Chloride,Year2,Week48,n=598: number analyzed (Participants) | 598
  Chloride,Year2,Week48,n=598 | 0.5 (2.81)
  Chloride,Year3,Week24,n=535: number analyzed (Participants) | 535
  Chloride,Year3,Week24,n=535 | 0.7 (3.04)
  Chloride,Year3,Week48,n=488: number analyzed (Participants) | 488
  Chloride,Year3,Week48,n=488 | 0.6 (2.73)
  Chloride,Year4,Week24,n=439: number analyzed (Participants) | 439
  Chloride,Year4,Week24,n=439 | 0.5 (2.74)
  Chloride,Year4,Week48,n=421: number analyzed (Participants) | 421
  Chloride,Year4,Week48,n=421 | 0.7 (2.84)
  Chloride,Year5,Week24,n=392: number analyzed (Participants) | 392
  Chloride,Year5,Week24,n=392 | 0.6 (2.95)
  Chloride,Year5,Week48,n=362: number analyzed (Participants) | 362
  Chloride,Year5,Week48,n=362 | 0.6 (2.77)
  Chloride,Year6,Week24,n=304: number analyzed (Participants) | 304
  Chloride,Year6,Week24,n=304 | 1.0 (2.74)
  Chloride,Year6,Week48,n=286: number analyzed (Participants) | 286
  Chloride,Year6,Week48,n=286 | 0.8 (2.67)
  Chloride,Year7,Week24,n=183: number analyzed (Participants) | 183
  Chloride,Year7,Week24,n=183 | 0.7 (2.57)
  Chloride,Year7,Week48,n=130: number analyzed (Participants) | 130
  Chloride,Year7,Week48,n=130 | 1.1 (2.73)
  Chloride,Year8,Week24,n=52: number analyzed (Participants) | 52
  Chloride,Year8,Week24,n=52 | 1.3 (2.86)
  Chloride,Year8,Week48,n=13: number analyzed (Participants) | 13
  Chloride,Year8,Week48,n=13 | 1.2 (3.54)
  Chloride,Year9,Week24,n=6: number analyzed (Participants) | 6
  Chloride,Year9,Week24,n=6 | 3.2 (1.47)
  Chloride,Year9,Week48,n=1: number analyzed (Participants) | 1
  Chloride,Year9,Week48,n=1 | 1.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Chloride,Exit,n=624: number analyzed (Participants) | 624
  Chloride,Exit,n=624 | 0.4 (3.06)
  Chloride,8 Week Follow up,n=538: number analyzed (Participants) | 538
  Chloride,8 Week Follow up,n=538 | 0.4 (2.82)
  Mg,Year1,Week4,n=707: number analyzed (Participants) | 707
  Mg,Year1,Week4,n=707 | -0.003 (0.0583)
  Mg,Year1,Week 12,n=705: number analyzed (Participants) | 705
  Mg,Year1,Week 12,n=705 | -0.006 (0.0647)
  Mg,Year1,Week 24,n=703: number analyzed (Participants) | 703
  Mg,Year1,Week 24,n=703 | -0.003 (0.0604)
  Mg,Year1,Week 36,n=684: number analyzed (Participants) | 684
  Mg,Year1,Week 36,n=684 | -0.004 (0.0616)
  Mg,Year1,Week 48,n=693: number analyzed (Participants) | 693
  Mg,Year1,Week 48,n=693 | 0.002 (0.0597)
  Mg,Year2,Week 24,n=643: number analyzed (Participants) | 643
  Mg,Year2,Week 24,n=643 | 0.002 (0.0694)
  Mg,Year2,Week 48,n=598: number analyzed (Participants) | 598
  Mg,Year2,Week 48,n=598 | 0.001 (0.0711)
  Mg,Year3,Week 24,n=535: number analyzed (Participants) | 535
  Mg,Year3,Week 24,n=535 | 0.010 (0.0668)
  Mg,Year3,Week 48,n=488: number analyzed (Participants) | 488
  Mg,Year3,Week 48,n=488 | 0.010 (0.0669)
  Mg,Year4,Week 24,n=439: number analyzed (Participants) | 439
  Mg,Year4,Week 24,n=439 | 0.016 (0.0700)
  Mg,Year4,Week 48,n=421: number analyzed (Participants) | 421
  Mg,Year4,Week 48,n=421 | 0.017 (0.0709)
  Mg,Year 5,Week 24,n=393: number analyzed (Participants) | 393
  Mg,Year 5,Week 24,n=393 | 0.016 (0.0673)
  Mg,Year 5,Week 48,n=362: number analyzed (Participants) | 362
  Mg,Year 5,Week 48,n=362 | 0.021 (0.0688)
  Mg,Year 6,Week 24,n=304: number analyzed (Participants) | 304
  Mg,Year 6,Week 24,n=304 | 0.013 (0.0718)
  Mg,Year 6,Week 48,n=286: number analyzed (Participants) | 286
  Mg,Year 6,Week 48,n=286 | 0.011 (0.0639)
  Mg,Year 7,Week 24,n=183: number analyzed (Participants) | 183
  Mg,Year 7,Week 24,n=183 | 0.010 (0.0692)
  Mg,Year 7,Week 48,n=130: number analyzed (Participants) | 130
  Mg,Year 7,Week 48,n=130 | 0.013 (0.0635)
  Mg,Year 8,Week 24,n=52: number analyzed (Participants) | 52
  Mg,Year 8,Week 24,n=52 | 0.025 (0.0702)
  Mg,Year 8,Week 48,n=13: number analyzed (Participants) | 13
  Mg,Year 8,Week 48,n=13 | 0.042 (0.0685)
  Mg,Year 9,Week 24,n=6: number analyzed (Participants) | 6
  Mg,Year 9,Week 24,n=6 | 0.030 (0.0613)
  Mg,Year 9,Week 48,n=1: number analyzed (Participants) | 1
  Mg,Year 9,Week 48,n=1 | 0.040 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Mg, Exit,n=625: number analyzed (Participants) | 625
  Mg, Exit,n=625 | 0.022 (0.0738)
  Mg,8 Week Follow up,n=539: number analyzed (Participants) | 539
  Mg,8 Week Follow up,n=539 | 0.021 (0.0729)
  Phos, Year1, Week4,n=707: number analyzed (Participants) | 707
  Phos, Year1, Week4,n=707 | 0.0102 (0.1908)
  Phos, Year1, Week12,n=705: number analyzed (Participants) | 705
  Phos, Year1, Week12,n=705 | 0.0004 (0.1999)
  Phos, Year1, Week24,n=703: number analyzed (Participants) | 703
  Phos, Year1, Week24,n=703 | -0.0126 (0.1964)
  Phos, Year1, Week 36,n=684: number analyzed (Participants) | 684
  Phos, Year1, Week 36,n=684 | 0.0101 (0.1976)
  Phos, Year1, Week48,n=693: number analyzed (Participants) | 693
  Phos, Year1, Week48,n=693 | -0.0110 (0.2086)
  Phos, Year2, Week24,n=643: number analyzed (Participants) | 643
  Phos, Year2, Week24,n=643 | -0.0026 (0.2138)
  Phos, Year2, Week48,n=598: number analyzed (Participants) | 598
  Phos, Year2, Week48,n=598 | -0.0044 (0.2062)
  Phos, Year3, Week24,n=535: number analyzed (Participants) | 535
  Phos, Year3, Week24,n=535 | -0.0109 (0.2028)
  Phos, Year3, Week48,n=488: number analyzed (Participants) | 488
  Phos, Year3, Week48,n=488 | -0.0185 (0.2138)
  Phos, Year4, Week24,n=439: number analyzed (Participants) | 439
  Phos, Year4, Week24,n=439 | -0.0072 (0.2067)
  Phos, Year4, Week48,n=421: number analyzed (Participants) | 421
  Phos, Year4, Week48,n=421 | -0.0143 (0.2118)
  Phos, Year5, Week24,n=393: number analyzed (Participants) | 393
  Phos, Year5, Week24,n=393 | -0.0199 (0.2751)
  Phos, Year5, Week48,n=362: number analyzed (Participants) | 362
  Phos, Year5, Week48,n=362 | -0.0320 (0.2145)
  Phos, Year6, Week24,n=304: number analyzed (Participants) | 304
  Phos, Year6, Week24,n=304 | -0.0238 (0.2214)
  Phos, Year6, Week48,n=286: number analyzed (Participants) | 286
  Phos, Year6, Week48,n=286 | -0.0123 (0.2113)
  Phos, Year 7, Week 24,n=183: number analyzed (Participants) | 183
  Phos, Year 7, Week 24,n=183 | -0.0196 (0.1970)
  Phos, Year 7, Week 48,n=130: number analyzed (Participants) | 130
  Phos, Year 7, Week 48,n=130 | -0.0101 (0.1912)
  Phos, Year 8, Week 24,n=52: number analyzed (Participants) | 52
  Phos, Year 8, Week 24,n=52 | -0.0041 (0.2038)
  Phos, Year 8, Week48,n=13: number analyzed (Participants) | 13
  Phos, Year 8, Week48,n=13 | -0.0340 (0.1337)
  Phos, Year9, Week 24,n=6: number analyzed (Participants) | 6
  Phos, Year9, Week 24,n=6 | -0.0803 (0.0823)
  Phos, Year 9, Week 48,n=1: number analyzed (Participants) | 1
  Phos, Year 9, Week 48,n=1 | 0.0447 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Phos, Exit, n=625: number analyzed (Participants) | 625
  Phos, Exit, n=625 | -0.0111 (0.2243)
  Phos, 8 Week Follow up,n=539: number analyzed (Participants) | 539
  Phos, 8 Week Follow up,n=539 | -0.0034 (0.2233)
  K, Year 1, Week 4, n=701: number analyzed (Participants) | 701
  K, Year 1, Week 4, n=701 | 0.07 (0.411)
  K, Year 1, Week 12, n=700: number analyzed (Participants) | 700
  K, Year 1, Week 12, n=700 | 0.03 (0.380)
  K, Year 1, Week 24, n=701: number analyzed (Participants) | 701
  K, Year 1, Week 24, n=701 | 0.01 (0.377)
  K, Year 1, Week 36, n=682: number analyzed (Participants) | 682
  K, Year 1, Week 36, n=682 | 0.04 (0.387)
  K, Year 1, Week 48, n=692: number analyzed (Participants) | 692
  K, Year 1, Week 48, n=692 | 0.01 (0.377)
  K, Year 2, Week 24, n=641: number analyzed (Participants) | 641
  K, Year 2, Week 24, n=641 | 0.01 (0.393)
  K, Year 2, Week 48, n=592: number analyzed (Participants) | 592
  K, Year 2, Week 48, n=592 | 0.02 (0.372)
  K, Year 3, Week 24, n=531: number analyzed (Participants) | 531
  K, Year 3, Week 24, n=531 | 0.05 (0.401)
  K, Year 3, Week 48, n=486: number analyzed (Participants) | 486
  K, Year 3, Week 48, n=486 | 0.06 (0.421)
  K, Year 4, Week 24, n=438: number analyzed (Participants) | 438
  K, Year 4, Week 24, n=438 | 0.06 (0.408)
  K, Year 4, Week 48, n=418: number analyzed (Participants) | 418
  K, Year 4, Week 48, n=418 | 0.03 (0.397)
  K, Year 5, Week 24, n=393: number analyzed (Participants) | 393
  K, Year 5, Week 24, n=393 | 0.08 (0.427)
  K, Year 5, Week 48, n=362: number analyzed (Participants) | 362
  K, Year 5, Week 48, n=362 | 0.02 (0.404)
  K, Year 6, Week 24, n=303: number analyzed (Participants) | 303
  K, Year 6, Week 24, n=303 | 0.06 (0.429)
  K, Year 6, Week 48, n=284: number analyzed (Participants) | 284
  K, Year 6, Week 48, n=284 | 0.05 (0.437)
  K, Year 7, Week 24, n=182: number analyzed (Participants) | 182
  K, Year 7, Week 24, n=182 | 0.05 (0.445)
  K, Year 7, Week 48, n=130: number analyzed (Participants) | 130
  K, Year 7, Week 48, n=130 | 0.05 (0.413)
  K, Year 8, Week 24, n=52: number analyzed (Participants) | 52
  K, Year 8, Week 24, n=52 | -0.02 (0.418)
  K, Year 8, Week 48, n=13: number analyzed (Participants) | 13
  K, Year 8, Week 48, n=13 | -0.12 (0.300)
  K, Year 9, Week 24, n=6: number analyzed (Participants) | 6
  K, Year 9, Week 24, n=6 | 0.05 (0.259)
  K, Year 9, Week 48, n=1: number analyzed (Participants) | 1
  K, Year 9, Week 48, n=1 | 0.00 (NA) — NA indicates standard deviation was not calculable for a single data point.
  K, Exit, n=624: number analyzed (Participants) | 624
  K, Exit, n=624 | 0.06 (0.435)
  K, 8 Week Follow up, n=537: number analyzed (Participants) | 537
  K, 8 Week Follow up, n=537 | 0.07 (0.452)
  Na, Year 1, Week 4, n=707: number analyzed (Participants) | 707
  Na, Year 1, Week 4, n=707 | 0.1 (2.07)
  Na, Year 1, Week 12, n=705: number analyzed (Participants) | 705
  Na, Year 1, Week 12, n=705 | 0.3 (2.25)
  Na, Year 1, Week 24, n=703: number analyzed (Participants) | 703
  Na, Year 1, Week 24, n=703 | 0.4 (2.16)
  Na, Year 1, Week 36, n=684: number analyzed (Participants) | 684
  Na, Year 1, Week 36, n=684 | 0.4 (2.10)
  Na, Year 1, Week 48, n=693: number analyzed (Participants) | 693
  Na, Year 1, Week 48, n=693 | 0.1 (2.09)
  Na, Year 2, Week 24, n=643: number analyzed (Participants) | 643
  Na, Year 2, Week 24, n=643 | -0.0 (2.30)
  Na, Year 2, Week 48, n=598: number analyzed (Participants) | 598
  Na, Year 2, Week 48, n=598 | 0.1 (2.63)
  Na, Year 3, Week 24, n=535: number analyzed (Participants) | 535
  Na, Year 3, Week 24, n=535 | 0.2 (2.54)
  Na, Year 3, Week 48, n=488: number analyzed (Participants) | 488
  Na, Year 3, Week 48, n=488 | 0.3 (2.36)
  Na, Year 4, Week 24, n=439: number analyzed (Participants) | 439
  Na, Year 4, Week 24, n=439 | 0.1 (2.31)
  Na, Year 4, Week 48, n=421: number analyzed (Participants) | 421
  Na, Year 4, Week 48, n=421 | 0.3 (2.36)
  Na, Year 5, Week 24, n=393: number analyzed (Participants) | 393
  Na, Year 5, Week 24, n=393 | 0.3 (2.61)
  Na, Year 5, Week 48, n=362: number analyzed (Participants) | 362
  Na, Year 5, Week 48, n=362 | 0.3 (2.18)
  Na, Year 6, Week 24, n=304: number analyzed (Participants) | 304
  Na, Year 6, Week 24, n=304 | 0.3 (2.22)
  Na, Year 6, Week 48, n=286: number analyzed (Participants) | 286
  Na, Year 6, Week 48, n=286 | 0.4 (2.44)
  Na, Year 7, Week 24, n=183: number analyzed (Participants) | 183
  Na, Year 7, Week 24, n=183 | 0.1 (2.22)
  Na, Year 7, Week 48, n=130: number analyzed (Participants) | 130
  Na, Year 7, Week 48, n=130 | 0.1 (2.38)
  Na, Year 8, Week 24, n=52: number analyzed (Participants) | 52
  Na, Year 8, Week 24, n=52 | 0.2 (2.67)
  Na, Year 8, Week 48, n=13: number analyzed (Participants) | 13
  Na, Year 8, Week 48, n=13 | 0.1 (2.14)
  Na, Year 9, Week 24, n=6: number analyzed (Participants) | 6
  Na, Year 9, Week 24, n=6 | 1.0 (1.79)
  Na, Year 9, Week 48, n=1: number analyzed (Participants) | 1
  Na, Year 9, Week 48, n=1 | -3.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Na, Exist, n=624: number analyzed (Participants) | 624
  Na, Exist, n=624 | 0.1 (2.55)
  Na, 8 Week Follow up, n=538: number analyzed (Participants) | 538
  Na, 8 Week Follow up, n=538 | 0.3 (2.36)

11. Primary Outcome: Change From Baseline in Blood Urea Nitrogen/Creatinine (BUN/Cr) at the Indicated Time Points
Description: Other chemistries parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 other chemistries parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in BUN/Cr is summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Ratio
  BUN/Cr,Year1,Week4,n=707: number analyzed (Participants) | 707
  BUN/Cr,Year1,Week4,n=707 | -0.2 (4.66)
  BUN/Cr,Year1,Week12,n=705: number analyzed (Participants) | 705
  BUN/Cr,Year1,Week12,n=705 | -0.3 (4.88)
  BUN/CrYear1,Week24,n=703: number analyzed (Participants) | 703
  BUN/CrYear1,Week24,n=703 | -0.7 (5.02)
  BUN/Cr,Year1,Week36,n=683: number analyzed (Participants) | 683
  BUN/Cr,Year1,Week36,n=683 | -0.5 (5.61)
  BUN/Cr,Year1,Week48,n=693: number analyzed (Participants) | 693
  BUN/Cr,Year1,Week48,n=693 | -0.2 (5.26)
  BUN/Cr,Year2,Week24,n=643: number analyzed (Participants) | 643
  BUN/Cr,Year2,Week24,n=643 | -0.1 (5.68)
  BUN/Cr,Year2,Week48,n=598: number analyzed (Participants) | 598
  BUN/Cr,Year2,Week48,n=598 | 0.5 (5.55)
  BUN/Cr,Year3,Week24,n=535: number analyzed (Participants) | 535
  BUN/Cr,Year3,Week24,n=535 | 1.4 (5.48)
  BUN/Cr,Year3,Week48,n=488: number analyzed (Participants) | 488
  BUN/Cr,Year3,Week48,n=488 | 1.2 (5.92)
  BUN/Cr,Year4,Week24,n=439: number analyzed (Participants) | 439
  BUN/Cr,Year4,Week24,n=439 | 1.4 (5.65)
  BUN/Cr,Year 4,Week48,n=421: number analyzed (Participants) | 421
  BUN/Cr,Year 4,Week48,n=421 | 1.0 (5.85)
  BUN/Cr,Year5,Week24,n=393: number analyzed (Participants) | 393
  BUN/Cr,Year5,Week24,n=393 | 0.7 (5.51)
  BUN/Cr,Year5,Week48,n=362: number analyzed (Participants) | 362
  BUN/Cr,Year5,Week48,n=362 | 1.0 (5.62)
  BUN/Cr,Year6,Week24,n=304: number analyzed (Participants) | 304
  BUN/Cr,Year6,Week24,n=304 | 1.0 (5.35)
  BUN/Cr,Year6,Week48,n=286: number analyzed (Participants) | 286
  BUN/Cr,Year6,Week48,n=286 | 1.3 (5.74)
  BUN/Cr,Year7,Week24,n=183: number analyzed (Participants) | 183
  BUN/Cr,Year7,Week24,n=183 | 0.8 (5.68)
  BUN/Cr,Year7,Week48,n=130: number analyzed (Participants) | 130
  BUN/Cr,Year7,Week48,n=130 | 1.2 (5.47)
  BUN/Cr,Year8,Week24,n=52: number analyzed (Participants) | 52
  BUN/Cr,Year8,Week24,n=52 | 3.3 (4.64)
  BUN/Cr,Year8,Week48,n=13: number analyzed (Participants) | 13
  BUN/Cr,Year8,Week48,n=13 | 3.5 (6.04)
  BUN/Cr,Year9,Week24,n=6: number analyzed (Participants) | 6
  BUN/Cr,Year9,Week24,n=6 | 3.5 (3.08)
  BUN/Cr,Year9,Week48,n=1: number analyzed (Participants) | 1
  BUN/Cr,Year9,Week48,n=1 | 1 (2.0)
  BUN/Cr,Exit,n=625: number analyzed (Participants) | 625
  BUN/Cr,Exit,n=625 | 0.9 (6.05)
  BUN/Cr,8 Week Follow up,n=539: number analyzed (Participants) | 539
  BUN/Cr,8 Week Follow up,n=539 | 0.9 (5.91)

12. Primary Outcome: Change From Baseline in Albumin (Alb) and Protein (Pro) at the Indicated Time Points
Description: Other chemistries parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 other chemistries parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Alb and Protein were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Grams per liter (g/L)
  Alb,Year1,Week4,n=707: number analyzed (Participants) | 707
  Alb,Year1,Week4,n=707 | -0.1 (2.36)
  Alb,Year1,Week12,n=705: number analyzed (Participants) | 705
  Alb,Year1,Week12,n=705 | 0.2 (2.67)
  Alb,Year1,Week24,n=703: number analyzed (Participants) | 703
  Alb,Year1,Week24,n=703 | 0.6 (3.03)
  Alb,Year1,Week36,n=684: number analyzed (Participants) | 684
  Alb,Year1,Week36,n=684 | 0.7 (3.23)
  Alb,Year1,Week48,n=693: number analyzed (Participants) | 693
  Alb,Year1,Week48,n=693 | 1.2 (3.52)
  Alb,Year2,Week24,n=643: number analyzed (Participants) | 643
  Alb,Year2,Week24,n=643 | 1.2 (3.49)
  Alb,Year2,Week48,n=598: number analyzed (Participants) | 598
  Alb,Year2,Week48,n=598 | 1.2 (3.67)
  Alb,Year3,Week24,n=535: number analyzed (Participants) | 535
  Alb,Year3,Week24,n=535 | 1.2 (3.78)
  Alb,Year3,Week48,n=488: number analyzed (Participants) | 488
  Alb,Year3,Week48,n=488 | 1.4 (4.02)
  Alb,Year4,Week24,n=439: number analyzed (Participants) | 439
  Alb,Year4,Week24,n=439 | 1.7 (4.02)
  Alb,Year 4,Week48,n=421: number analyzed (Participants) | 421
  Alb,Year 4,Week48,n=421 | 1.9 (4.04)
  Alb,Year5,Week24,n=393: number analyzed (Participants) | 393
  Alb,Year5,Week24,n=393 | 1.9 (3.85)
  Alb,Year5,Week48,n=362: number analyzed (Participants) | 362
  Alb,Year5,Week48,n=362 | 2.3 (3.89)
  Alb,Year6,Week24,n=304: number analyzed (Participants) | 304
  Alb,Year6,Week24,n=304 | 2.2 (3.78)
  Alb,Year6,Week48,n=286: number analyzed (Participants) | 286
  Alb,Year6,Week48,n=286 | 2.1 (4.07)
  Alb,Year7,Week24,n=183: number analyzed (Participants) | 183
  Alb,Year7,Week24,n=183 | 2.0 (3.60)
  Alb,Year7,Week48,n=130: number analyzed (Participants) | 130
  Alb,Year7,Week48,n=130 | 2.3 (3.92)
  Alb,Year8,Week24,n=52: number analyzed (Participants) | 52
  Alb,Year8,Week24,n=52 | 1.9 (4.16)
  Alb,Year8,Week48,n=13: number analyzed (Participants) | 13
  Alb,Year8,Week48,n=13 | 1.1 (4.11)
  Alb,Year9,Week24,n=6: number analyzed (Participants) | 6
  Alb,Year9,Week24,n=6 | 0.7 (3.01)
  Alb,Year9,Week48,n=1: number analyzed (Participants) | 1
  Alb,Year9,Week48,n=1 | 1.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Alb,Exit,n=625: number analyzed (Participants) | 625
  Alb,Exit,n=625 | 1.8 (4.74)
  Alb,8 Week Follow up,n=539: number analyzed (Participants) | 539
  Alb,8 Week Follow up,n=539 | 1.7 (4.66)
  Pro,Year1,Week4,n=707: number analyzed (Participants) | 707
  Pro,Year1,Week4,n=707 | -1.4 (3.81)
  Pro,Year1,Week12,n=705: number analyzed (Participants) | 705
  Pro,Year1,Week12,n=705 | -2.0 (4.30)
  Pro,Year1,Week24,n=703: number analyzed (Participants) | 703
  Pro,Year1,Week24,n=703 | -1.9 (4.68)
  Pro,Year1,Week36,n=684: number analyzed (Participants) | 684
  Pro,Year1,Week36,n=684 | -2.3 (4.75)
  Pro,Year1,Week48,n=693: number analyzed (Participants) | 693
  Pro,Year1,Week48,n=693 | -1.8 (4.94)
  Pro,Year2,Week24,n=643: number analyzed (Participants) | 643
  Pro,Year2,Week24,n=643 | -2.3 (5.05)
  Pro,Year2,Week48,n=598: number analyzed (Participants) | 598
  Pro,Year2,Week48,n=598 | -2.7 (5.53)
  Pro,Year3,Week24,n=535: number analyzed (Participants) | 535
  Pro,Year3,Week24,n=535 | -3.1 (5.62)
  Pro,Year3,Week48,n=488: number analyzed (Participants) | 488
  Pro,Year3,Week48,n=488 | -3.5 (5.91)
  Pro,Year4,Week24,n=439: number analyzed (Participants) | 439
  Pro,Year4,Week24,n=439 | -3.2 (5.87)
  Pro,Year 4,Week48,n=421: number analyzed (Participants) | 421
  Pro,Year 4,Week48,n=421 | -3.2 (6.07)
  Pro,Year5,Week24,n=393: number analyzed (Participants) | 393
  Pro,Year5,Week24,n=393 | -3.5 (5.75)
  Pro,Year5,Week48,n=362: number analyzed (Participants) | 362
  Pro,Year5,Week48,n=362 | -3.6 (5.78)
  Pro,Year6,Week24,n=304: number analyzed (Participants) | 304
  Pro,Year6,Week24,n=304 | -3.9 (5.57)
  Pro,Year6,Week48,n=286: number analyzed (Participants) | 286
  Pro,Year6,Week48,n=286 | -4.0 (5.79)
  Pro,Year7,Week24,n=183: number analyzed (Participants) | 183
  Pro,Year7,Week24,n=183 | -4.3 (5.36)
  Pro,Year7,Week48,n=130: number analyzed (Participants) | 130
  Pro,Year7,Week48,n=130 | -3.9 (5.32)
  Pro,Year8,Week24,n=52: number analyzed (Participants) | 52
  Pro,Year8,Week24,n=52 | -5.1 (6.38)
  Pro,Year8,Week48,n=13: number analyzed (Participants) | 13
  Pro,Year8,Week48,n=13 | -4.8 (5.02)
  Pro,Year9,Week24,n=6: number analyzed (Participants) | 6
  Pro,Year9,Week24,n=6 | -7.7 (7.03)
  Pro,Year9,Week48,n=1: number analyzed (Participants) | 1
  Pro,Year9,Week48,n=1 | 0.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Pro,Exit,n=625: number analyzed (Participants) | 625
  Pro,Exit,n=625 | -3.4 (6.45)
  Pro,8 Week Follow up,n=539: number analyzed (Participants) | 539
  Pro,8 Week Follow up,n=539 | -3.7 (6.42)

13. Primary Outcome: Change From Baseline in BUN and Glucose at the Indicated Time Points
Description: Other chemistries parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 other chemistries were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in BUN and Glucose were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
mmol/L
  BUN,Year1,Week4,n=707: number analyzed (Participants) | 707
  BUN,Year1,Week4,n=707 | 0.0299 (1.6783)
  BUN,Year1,Week12,n=705: number analyzed (Participants) | 705
  BUN,Year1,Week12,n=705 | 0.0402 (1.9768)
  BUN,Year1,Week24,n=703: number analyzed (Participants) | 703
  BUN,Year1,Week24,n=703 | -0.1443 (1.3723)
  BUN,Year1,Week36,n=683: number analyzed (Participants) | 683
  BUN,Year1,Week36,n=683 | -0.0592 (1.6916)
  BUN,Year1,Week48,n=693: number analyzed (Participants) | 693
  BUN,Year1,Week48,n=693 | -0.0406 (1.5541)
  BUN,Year2,Week24,n=643: number analyzed (Participants) | 643
  BUN,Year2,Week24,n=643 | -0.0760 (1.6652)
  BUN,Year2,Week48,n=598: number analyzed (Participants) | 598
  BUN,Year2,Week48,n=598 | 0.0631 (1.6429)
  BUN,Year3,Week24,n=535: number analyzed (Participants) | 535
  BUN,Year3,Week24,n=535 | 0.0524 (1.6850)
  BUN,Year3,Week48,n=488: number analyzed (Participants) | 488
  BUN,Year3,Week48,n=488 | -0.1013 (1.6910)
  BUN,Year4,Week24,n=439: number analyzed (Participants) | 439
  BUN,Year4,Week24,n=439 | 0.0967 (1.9398)
  BUN,Year 4,Week48,n=421: number analyzed (Participants) | 421
  BUN,Year 4,Week48,n=421 | 0.0672 (2.1393)
  BUN,Year5,Week24,n=393: number analyzed (Participants) | 393
  BUN,Year5,Week24,n=393 | -0.0291 (2.0169)
  BUN,Year5,Week48,n=362: number analyzed (Participants) | 362
  BUN,Year5,Week48,n=362 | 0.0899 (2.0903)
  BUN,Year6,Week24,n=304: number analyzed (Participants) | 304
  BUN,Year6,Week24,n=304 | 0.0959 (1.9852)
  BUN,Year6,Week48,n=286: number analyzed (Participants) | 286
  BUN,Year6,Week48,n=286 | 0.2325 (2.2724)
  BUN,Year7,Week24,n=183: number analyzed (Participants) | 183
  BUN,Year7,Week24,n=183 | -0.0026 (1.6623)
  BUN,Year7,Week48,n=130: number analyzed (Participants) | 130
  BUN,Year7,Week48,n=130 | 0.1455 (1.7145)
  BUN,Year8,Week24,n=52: number analyzed (Participants) | 52
  BUN,Year8,Week24,n=52 | 0.5458 (1.7299)
  BUN,Year8,Week48,n=13: number analyzed (Participants) | 13
  BUN,Year8,Week48,n=13 | 0.3883 (1.4603)
  BUN,Year9,Week24,n=6: number analyzed (Participants) | 6
  BUN,Year9,Week24,n=6 | 0.1648 (1.0466)
  BUN,Year9,Week48,n=1: number analyzed (Participants) | 1
  BUN,Year9,Week48,n=1 | 0.5700 (NA) — NA indicates standard deviation was not calculable for a single data point.
  BUN,Exit,n=625: number analyzed (Participants) | 625
  BUN,Exit,n=625 | 0.2448 (2.4618)
  BUN,8 Week Follow up,n=539: number analyzed (Participants) | 539
  BUN,8 Week Follow up,n=539 | 0.0822 (2.5567)
  Glucose,Year1,Week4,n=707: number analyzed (Participants) | 707
  Glucose,Year1,Week4,n=707 | -0.0031 (1.0221)
  Glucose,Year1,Week12,n=705: number analyzed (Participants) | 705
  Glucose,Year1,Week12,n=705 | 0.0333 (1.0627)
  Glucose,Year1,Week24,n=702: number analyzed (Participants) | 702
  Glucose,Year1,Week24,n=702 | -0.0396 (1.2656)
  Glucose,Year1,Week36,n=684: number analyzed (Participants) | 684
  Glucose,Year1,Week36,n=684 | 0.0099 (1.0269)
  Glucose,Year1,Week48,n=693: number analyzed (Participants) | 693
  Glucose,Year1,Week48,n=693 | 0.0010 (1.1726)
  Glucose,Year2,Week24,n=643: number analyzed (Participants) | 643
  Glucose,Year2,Week24,n=643 | 0.0143 (1.3227)
  Glucose,Year2,Week48,n=598: number analyzed (Participants) | 598
  Glucose,Year2,Week48,n=598 | -0.0082 (1.1352)
  Glucose,Year3,Week24,n=535: number analyzed (Participants) | 535
  Glucose,Year3,Week24,n=535 | -0.0159 (1.3222)
  Glucose,Year3,Week48,n=488: number analyzed (Participants) | 488
  Glucose,Year3,Week48,n=488 | 0.0309 (1.1841)
  Glucose,Year4,Week24,n=439: number analyzed (Participants) | 439
  Glucose,Year4,Week24,n=439 | -0.0160 (1.2213)
  Glucose,Year 4,Week48,n=421: number analyzed (Participants) | 421
  Glucose,Year 4,Week48,n=421 | -0.0259 (1.1936)
  Glucose,Year5,Week24,n=393: number analyzed (Participants) | 393
  Glucose,Year5,Week24,n=393 | 0.0554 (1.1255)
  Glucose,Year5,Week48,n=362: number analyzed (Participants) | 362
  Glucose,Year5,Week48,n=362 | 0.0655 (1.2946)
  Glucose,Year6,Week24,n=303: number analyzed (Participants) | 303
  Glucose,Year6,Week24,n=303 | 0.1290 (1.1163)
  Glucose,Year6,Week48,n=286: number analyzed (Participants) | 286
  Glucose,Year6,Week48,n=286 | 0.2001 (1.2411)
  Glucose,Year7,Week24,n=183: number analyzed (Participants) | 183
  Glucose,Year7,Week24,n=183 | 0.2303 (1.0514)
  Glucose,Year7,Week48,n=130: number analyzed (Participants) | 130
  Glucose,Year7,Week48,n=130 | 0.2335 (0.8346)
  Glucose,Year8,Week24,n=52: number analyzed (Participants) | 52
  Glucose,Year8,Week24,n=52 | 0.3301 (0.9052)
  Glucose,Year8,Week48,n=13: number analyzed (Participants) | 13
  Glucose,Year8,Week48,n=13 | 0.1431 (0.8115)
  Glucose,Year9,Week24,n=6: number analyzed (Participants) | 6
  Glucose,Year9,Week24,n=6 | 0.2128 (0.4914)
  Glucose,Year9,Week48,n=1: number analyzed (Participants) | 1
  Glucose,Year9,Week48,n=1 | 0.4739 (NA) — NA indicates standard deviation was not calculable for a single data point
  Glucose,Exit,n=624: number analyzed (Participants) | 624
  Glucose,Exit,n=624 | 0.1842 (1.8723)
  Glucose,8 Week Follow up,n=539: number analyzed (Participants) | 539
  Glucose,8 Week Follow up,n=539 | 0.0338 (1.4139)

14. Primary Outcome: Change From Baseline in Creatinine (Cr) and Urate at the Indicated Time Points
Description: Other chemistries parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 other chemistries were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Cr and Urate were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Micromoles per liter (µmol/L)
  Urate,Year1,Week4,n=707: number analyzed (Participants) | 707
  Urate,Year1,Week4,n=707 | 1.0332 (45.8504)
  Urate,Year1,Week12,n=704: number analyzed (Participants) | 704
  Urate,Year1,Week12,n=704 | 0.4089 (54.3182)
  Urate,Year1,Week24,n=703: number analyzed (Participants) | 703
  Urate,Year1,Week24,n=703 | -0.0510 (49.2328)
  Urate,Year1,Week36,n=684: number analyzed (Participants) | 684
  Urate,Year1,Week36,n=684 | 0.6713 (50.7341)
  Urate,Year1,Week48,n=693: number analyzed (Participants) | 693
  Urate,Year1,Week48,n=693 | -1.5147 (50.5928)
  Urate,Year2,Week24,n=643: number analyzed (Participants) | 643
  Urate,Year2,Week24,n=643 | 2.7246 (55.7467)
  Urate,Year2,Week48,n=598: number analyzed (Participants) | 598
  Urate,Year2,Week48,n=598 | 4.1255 (60.0251)
  Urate,Year3,Week24,n=535: number analyzed (Participants) | 535
  Urate,Year3,Week24,n=535 | 6.7497 (60.4118)
  Urate,Year3,Week48,n=488: number analyzed (Participants) | 488
  Urate,Year3,Week48,n=488 | 6.9744 (63.6876)
  Urate,Year4,Week24,n=439: number analyzed (Participants) | 439
  Urate,Year4,Week24,n=439 | 5.9658 (66.6167)
  Urate,Year 4,Week48,n=421: number analyzed (Participants) | 421
  Urate,Year 4,Week48,n=421 | 4.0772 (67.9587)
  Urate,Year5,Week24,n=393: number analyzed (Participants) | 393
  Urate,Year5,Week24,n=393 | -0.5634 (66.9130)
  Urate,Year5,Week48,n=362: number analyzed (Participants) | 362
  Urate,Year5,Week48,n=362 | -0.8979 (67.3843)
  Urate,Year6,Week24,n=304: number analyzed (Participants) | 304
  Urate,Year6,Week24,n=304 | 2.9530 (62.3168)
  Urate,Year6,Week48,n=286: number analyzed (Participants) | 286
  Urate,Year6,Week48,n=286 | 1.1244 (67.3175)
  Urate,Year7,Week24,n=183: number analyzed (Participants) | 183
  Urate,Year7,Week24,n=183 | 2.1521 (53.0854)
  Urate,Year7,Week48,n=130: number analyzed (Participants) | 130
  Urate,Year7,Week48,n=130 | 4.0062 (58.3577)
  Urate,Year8,Week24,n=52: number analyzed (Participants) | 52
  Urate,Year8,Week24,n=52 | -1.1003 (51.8840)
  Urate,Year8,Week48,n=13: number analyzed (Participants) | 13
  Urate,Year8,Week48,n=13 | 29.2043 (80.1811)
  Urate,Year9,Week24,n=6: number analyzed (Participants) | 6
  Urate,Year9,Week24,n=6 | 0.2187 (45.1947)
  Urate,Year9,Week48,n=1: number analyzed (Participants) | 1
  Urate,Year9,Week48,n=1 | -69.6640 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Urate,Exit,n=625: number analyzed (Participants) | 625
  Urate,Exit,n=625 | 1.6479 (74.4078)
  Urate,8 Week Follow up,n=539: number analyzed (Participants) | 539
  Urate,8 Week Follow up,n=539 | -2.7404 (75.5887)
  Cr,Year1,Week4,n=707: number analyzed (Participants) | 707
  Cr,Year1,Week4,n=707 | 0.913 (14.2222)
  Cr,Year1,Week12,n=705: number analyzed (Participants) | 705
  Cr,Year1,Week12,n=705 | 0.751 (14.0933)
  Cr,Year1,Week24,n=703: number analyzed (Participants) | 703
  Cr,Year1,Week24,n=703 | 0.823 (9.5372)
  Cr,Year1,Week36,n=684: number analyzed (Participants) | 684
  Cr,Year1,Week36,n=684 | 1.313 (13.1107)
  Cr,Year1,Week48,n=693: number analyzed (Participants) | 693
  Cr,Year1,Week48,n=693 | 0.439 (11.1364)
  Cr,Year2,Week24,n=643: number analyzed (Participants) | 643
  Cr,Year2,Week24,n=643 | -0.217 (13.9502)
  Cr,Year2,Week48,n=598: number analyzed (Participants) | 598
  Cr,Year2,Week48,n=598 | -0.922 (13.6541)
  Cr,Year3,Week24,n=535: number analyzed (Participants) | 535
  Cr,Year3,Week24,n=535 | -3.870 (17.8146)
  Cr,Year3,Week48,n=488: number analyzed (Participants) | 488
  Cr,Year3,Week48,n=488 | -4.844 (17.7059)
  Crea,Year4,Week24,n=439: number analyzed (Participants) | 439
  Crea,Year4,Week24,n=439 | -3.196 (22.2874)
  Crea,Year 4,Week48,n=421: number analyzed (Participants) | 421
  Crea,Year 4,Week48,n=421 | -2.145 (30.9370)
  Cr,Year5,Week24,n=393: number analyzed (Participants) | 393
  Cr,Year5,Week24,n=393 | -1.999 (32.6689)
  Cr,Year5,Week48,n=362: number analyzed (Participants) | 362
  Cr,Year5,Week48,n=362 | -1.918 (28.8788)
  Cr,Year6,Week24,n=304: number analyzed (Participants) | 304
  Cr,Year6,Week24,n=304 | -2.125 (24.2374)
  Cr,Year6,Week48,n=286: number analyzed (Participants) | 286
  Cr,Year6,Week48,n=286 | -1.534 (28.8012)
  Cr,Year7,Week24,n=183: number analyzed (Participants) | 183
  Cr,Year7,Week24,n=183 | -2.511 (15.6881)
  Cr,Year7,Week48,n=130: number analyzed (Participants) | 130
  Cr,Year7,Week48,n=130 | -2.586 (14.0864)
  Cr,Year8,Week24,n=52: number analyzed (Participants) | 52
  Cr,Year8,Week24,n=52 | -4.659 (16.3056)
  Cr,Year8,Week48,n=13: number analyzed (Participants) | 13
  Cr,Year8,Week48,n=13 | -6.175 (6.6311)
  Cr,Year9,Week24,n=6: number analyzed (Participants) | 6
  Cr,Year9,Week24,n=6 | -8.933 (5.6925)
  Cr,Year9,Week48,n=1: number analyzed (Participants) | 1
  Cr,Year9,Week48,n=1 | 0.040 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Cr,Exit,n=624: number analyzed (Participants) | 624
  Cr,Exit,n=624 | 0.606 (35.9813)
  Cr,8 Week Follow up,n=539: number analyzed (Participants) | 539
  Cr,8 Week Follow up,n=539 | -1.108 (39.0635)

15. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (GGT) and Lactate Dehydrogenase (LDH) Levels
Description: Liver function parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 liver function parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in ALT, ALP, AST, GGT and LDH were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: International Units/liter (IU/L)
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
International Units/liter (IU/L)
  ALT, Year 1 Week 4, n=707: number analyzed (Participants) | 707
  ALT, Year 1 Week 4, n=707 | -0.4 (10.18)
  ALT, Year 1 Week 12, n=705: number analyzed (Participants) | 705
  ALT, Year 1 Week 12, n=705 | -0.9 (12.31)
  ALT, Year 1 Week 24, n=703: number analyzed (Participants) | 703
  ALT, Year 1 Week 24, n=703 | -0.9 (19.46)
  ALT, Year 1 Week 36, n=684: number analyzed (Participants) | 684
  ALT, Year 1 Week 36, n=684 | -1.0 (15.61)
  ALT, Year 1 Week 48, n=693: number analyzed (Participants) | 693
  ALT, Year 1 Week 48, n=693 | -0.7 (15.04)
  ALT, Year 2 Week 24, n=643: number analyzed (Participants) | 643
  ALT, Year 2 Week 24, n=643 | 0.2 (23.56)
  ALT, Year 2 Week 48, n=598: number analyzed (Participants) | 598
  ALT, Year 2 Week 48, n=598 | 2.7 (57.67)
  ALT, Year 3 Week 24, n=535: number analyzed (Participants) | 535
  ALT, Year 3 Week 24, n=535 | -1.3 (14.40)
  ALT, Year 3 Week 48, n=488: number analyzed (Participants) | 488
  ALT, Year 3 Week 48, n=488 | 0.1 (21.21)
  ALT, Year 4 Week 24, n=439: number analyzed (Participants) | 439
  ALT, Year 4 Week 24, n=439 | -0.1 (18.72)
  ALT, Year 4 Week 48, n=421: number analyzed (Participants) | 421
  ALT, Year 4 Week 48, n=421 | -0.6 (17.59)
  ALT, Year 5 Week 24, n=393: number analyzed (Participants) | 393
  ALT, Year 5 Week 24, n=393 | -1.3 (18.74)
  ALT, Year 5 Week 48, n=362: number analyzed (Participants) | 362
  ALT, Year 5 Week 48, n=362 | -0.4 (22.72)
  ALT, Year 6 Week 24, n=304: number analyzed (Participants) | 304
  ALT, Year 6 Week 24, n=304 | -0.2 (20.54)
  ALT, Year 6 Week 48, n=286: number analyzed (Participants) | 286
  ALT, Year 6 Week 48, n=286 | 0.9 (20.94)
  ALT, Year 7 Week 24, n=183: number analyzed (Participants) | 183
  ALT, Year 7 Week 24, n=183 | 1.3 (19.46)
  ALT, Year 7 Week 48, n=130: number analyzed (Participants) | 130
  ALT, Year 7 Week 48, n=130 | -0.1 (16.79)
  ALT, Year 8 Week 24, n=52: number analyzed (Participants) | 52
  ALT, Year 8 Week 24, n=52 | 2.7 (31.15)
  ALT, Year 8 Week 48, n=13: number analyzed (Participants) | 13
  ALT, Year 8 Week 48, n=13 | 5.8 (33.54)
  ALT, Year 9 Week 24, n=6: number analyzed (Participants) | 6
  ALT, Year 9 Week 24, n=6 | 9.3 (27.77)
  ALT, Year 9 Week 48, n=1: number analyzed (Participants) | 1
  ALT, Year 9 Week 48, n=1 | -6.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  ALT, Exit, n=624: number analyzed (Participants) | 624
  ALT, Exit, n=624 | -0.6 (17.03)
  ALT, 8 Week follow-up, n=539: number analyzed (Participants) | 539
  ALT, 8 Week follow-up, n=539 | -0.8 (17.06)
  ALP, Year 1 Week 4, n=707: number analyzed (Participants) | 707
  ALP, Year 1 Week 4, n=707 | 0.0 (11.85)
  ALP, Year 1 Week 12, n=705: number analyzed (Participants) | 705
  ALP, Year 1 Week 12, n=705 | 0.5 (13.31)
  ALP, Year 1 Week 24, n=703: number analyzed (Participants) | 703
  ALP, Year 1 Week 24, n=703 | 2.1 (17.76)
  ALP, Year 1 Week 36, n=684: number analyzed (Participants) | 684
  ALP, Year 1 Week 36, n=684 | 1.7 (22.81)
  ALP, Year 1 Week 48, n=693: number analyzed (Participants) | 693
  ALP, Year 1 Week 48, n=693 | 4.6 (21.18)
  ALP, Year 2 Week 24, n=643: number analyzed (Participants) | 643
  ALP, Year 2 Week 24, n=643 | 5.1 (21.58)
  ALP, Year 2 Week 48, n=598: number analyzed (Participants) | 598
  ALP, Year 2 Week 48, n=598 | 6.1 (23.23)
  ALP, Year 3 Week 24, n=535: number analyzed (Participants) | 535
  ALP, Year 3 Week 24, n=535 | 5.9 (18.95)
  ALP, Year 3 Week 48, n=488: number analyzed (Participants) | 488
  ALP, Year 3 Week 48, n=488 | 7.3 (22.22)
  ALP, Year 4 Week 24, n=439: number analyzed (Participants) | 439
  ALP, Year 4 Week 24, n=439 | 7.2 (21.56)
  ALP, Year 4 Week 48, n=421: number analyzed (Participants) | 421
  ALP, Year 4 Week 48, n=421 | 8.1 (27.35)
  ALP, Year 5 Week 24, n=393: number analyzed (Participants) | 393
  ALP, Year 5 Week 24, n=393 | 7.2 (21.01)
  ALP, Year 5 Week 48, n=362: number analyzed (Participants) | 362
  ALP, Year 5 Week 48, n=362 | 8.5 (20.61)
  ALP, Year 6 Week 24, n=304: number analyzed (Participants) | 304
  ALP, Year 6 Week 24, n=304 | 9.4 (23.28)
  ALP, Year 6 Week 48, n=286: number analyzed (Participants) | 286
  ALP, Year 6 Week 48, n=286 | 11.5 (27.39)
  ALP, Year 7 Week 24, n=183: number analyzed (Participants) | 183
  ALP, Year 7 Week 24, n=183 | 10.9 (28.08)
  ALP, Year 7 Week 48, n=130: number analyzed (Participants) | 130
  ALP, Year 7 Week 48, n=130 | 7.5 (22.50)
  ALP, Year 8 Week 24, n=52: number analyzed (Participants) | 52
  ALP, Year 8 Week 24, n=52 | 12.9 (26.64)
  ALP, Year 8 Week 48, n=13: number analyzed (Participants) | 13
  ALP, Year 8 Week 48, n=13 | 6.1 (30.04)
  ALP, Year 9 Week 24, n=6: number analyzed (Participants) | 6
  ALP, Year 9 Week 24, n=6 | 4.2 (35.43)
  ALP, Year 9 Week 48, n=1: number analyzed (Participants) | 1
  ALP, Year 9 Week 48, n=1 | 12.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  ALP, Exit, n=625: number analyzed (Participants) | 625
  ALP, Exit, n=625 | 7.5 (25.35)
  ALP, 8 Week follow-up, n=539: number analyzed (Participants) | 539
  ALP, 8 Week follow-up, n=539 | 6.1 (23.00)
  AST, Year 1 Week 4, n=701: number analyzed (Participants) | 701
  AST, Year 1 Week 4, n=701 | -0.6 (10.56)
  AST, Year 1 Week 12, n=700: number analyzed (Participants) | 700
  AST, Year 1 Week 12, n=700 | -1.3 (14.12)
  AST, Year 1 Week 24, n=701: number analyzed (Participants) | 701
  AST, Year 1 Week 24, n=701 | -1.0 (20.79)
  AST, Year 1 Week 36, n=682: number analyzed (Participants) | 682
  AST, Year 1 Week 36, n=682 | -1.0 (17.88)
  AST, Year 1 Week 48, n=692: number analyzed (Participants) | 692
  AST, Year 1 Week 48, n=692 | -0.9 (14.38)
  AST, Year 2 Week 24, n=641: number analyzed (Participants) | 641
  AST, Year 2 Week 24, n=641 | -0.4 (22.22)
  AST, Year 2 Week 48, n=592: number analyzed (Participants) | 592
  AST, Year 2 Week 48, n=592 | 2.9 (57.25)
  AST, Year 3 Week 24, n=531: number analyzed (Participants) | 531
  AST, Year 3 Week 24, n=531 | -1.4 (13.26)
  AST, Year 3 Week 48, n=486: number analyzed (Participants) | 486
  AST, Year 3 Week 48, n=486 | -0.5 (17.23)
  AST, Year 4 Week 24, n=438: number analyzed (Participants) | 438
  AST, Year 4 Week 24, n=438 | -0.9 (14.60)
  AST, Year 4 Week 48, n=418: number analyzed (Participants) | 418
  AST, Year 4 Week 48, n=418 | -0.7 (15.32)
  AST, Year 5 Week 24, n=393: number analyzed (Participants) | 393
  AST, Year 5 Week 24, n=393 | -1.3 (16.07)
  AST, Year 5 Week 48, n=362: number analyzed (Participants) | 362
  AST, Year 5 Week 48, n=362 | -0.8 (18.57)
  AST, Year 6 Week 24, n=303: number analyzed (Participants) | 303
  AST, Year 6 Week 24, n=303 | -0.5 (16.95)
  AST, Year 6 Week 48, n=284: number analyzed (Participants) | 284
  AST, Year 6 Week 48, n=284 | -0.2 (19.00)
  AST, Year 7 Week 24, n=182: number analyzed (Participants) | 182
  AST, Year 7 Week 24, n=182 | 0.6 (13.43)
  AST, Year 7 Week 48, n=130: number analyzed (Participants) | 130
  AST, Year 7 Week 48, n=130 | -0.3 (10.78)
  AST, Year 8 Week 24, n=52: number analyzed (Participants) | 52
  AST, Year 8 Week 24, n=52 | 3.0 (33.93)
  AST, Year 8 Week 48, n=13: number analyzed (Participants) | 13
  AST, Year 8 Week 48, n=13 | 5.8 (24.01)
  AST, Year 9 Week 24, n=6: number analyzed (Participants) | 6
  AST, Year 9 Week 24, n=6 | 7.7 (19.63)
  AST, Year 9 Week 48, n=1: number analyzed (Participants) | 1
  AST, Year 9 Week 48, n=1 | 0.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  AST, Exit, n=625: number analyzed (Participants) | 625
  AST, Exit, n=625 | -0.6 (18.88)
  AST, 8 Week follow-up, n=539: number analyzed (Participants) | 539
  AST, 8 Week follow-up, n=539 | -1.1 (16.58)
  GGT, Year 1 Week 4, n=707: number analyzed (Participants) | 707
  GGT, Year 1 Week 4, n=707 | -0.4 (23.39)
  GGT, Year 1 Week 12, n=705: number analyzed (Participants) | 705
  GGT, Year 1 Week 12, n=705 | -1.4 (23.12)
  GGT, Year 1 Week 24, n=703: number analyzed (Participants) | 703
  GGT, Year 1 Week 24, n=703 | -0.2 (39.50)
  GGT, Year 1 Week 36, n=684: number analyzed (Participants) | 684
  GGT, Year 1 Week 36, n=684 | 1.0 (64.60)
  GGT, Year 1 Week 48, n=693: number analyzed (Participants) | 693
  GGT, Year 1 Week 48, n=693 | 0.9 (35.99)
  GGT, Year 2 Week 24, n=643: number analyzed (Participants) | 643
  GGT, Year 2 Week 24, n=643 | -0.7 (34.81)
  GGT, Year 2 Week 48, n=598: number analyzed (Participants) | 598
  GGT, Year 2 Week 48, n=598 | 0.1 (34.63)
  GGT, Year 3 Week 24, n=535: number analyzed (Participants) | 535
  GGT, Year 3 Week 24, n=535 | -1.6 (33.88)
  GGT, Year 3 Week 48, n=488: number analyzed (Participants) | 488
  GGT, Year 3 Week 48, n=488 | 1.7 (45.42)
  GGT, Year 4 Week 24, n=439: number analyzed (Participants) | 439
  GGT, Year 4 Week 24, n=439 | 0.1 (39.13)
  GGT, Year 4 Week 48, n=421: number analyzed (Participants) | 421
  GGT, Year 4 Week 48, n=421 | 1.1 (54.41)
  GGT, Year 5 Week 24, n=393: number analyzed (Participants) | 393
  GGT, Year 5 Week 24, n=393 | -2.0 (37.17)
  GGT, Year 5 Week 48, n=362: number analyzed (Participants) | 362
  GGT, Year 5 Week 48, n=362 | -0.7 (43.39)
  GGT, Year 6 Week 24, n=304: number analyzed (Participants) | 304
  GGT, Year 6 Week 24, n=304 | -1.0 (42.04)
  GGT, Year 6 Week 48, n=286: number analyzed (Participants) | 286
  GGT, Year 6 Week 48, n=286 | 1.3 (41.84)
  GGT, Year 7 Week 24, n=183: number analyzed (Participants) | 183
  GGT, Year 7 Week 24, n=183 | 1.8 (37.06)
  GGT, Year 7 Week 48, n=130: number analyzed (Participants) | 130
  GGT, Year 7 Week 48, n=130 | -1.0 (27.86)
  GGT, Year 8 Week 24, n=52: number analyzed (Participants) | 52
  GGT, Year 8 Week 24, n=52 | 2.7 (39.90)
  GGT, Year 8 Week 48, n=13: number analyzed (Participants) | 13
  GGT, Year 8 Week 48, n=13 | -0.3 (27.97)
  GGT, Year 9 Week 24, n=6: number analyzed (Participants) | 6
  GGT, Year 9 Week 24, n=6 | 13.3 (26.96)
  GGT, Year 9 Week 48, n=1: number analyzed (Participants) | 1
  GGT, Year 9 Week 48, n=1 | -7.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  GGT, Exit, n=625: number analyzed (Participants) | 625
  GGT, Exit, n=625 | 0.7 (41.40)
  GGT, 8 Week follow-up, n=539: number analyzed (Participants) | 539
  GGT, 8 Week follow-up, n=539 | 0.2 (39.22)
  LDH, Year 1 Week 4, n=701: number analyzed (Participants) | 701
  LDH, Year 1 Week 4, n=701 | -4.1 (77.93)
  LDH, Year 1 Week 12, n=700: number analyzed (Participants) | 700
  LDH, Year 1 Week 12, n=700 | -6.0 (80.55)
  LDH, Year 1 Week 24, n=701: number analyzed (Participants) | 701
  LDH, Year 1 Week 24, n=701 | -6.6 (80.09)
  LDH, Year 1 Week 36, n=682: number analyzed (Participants) | 682
  LDH, Year 1 Week 36, n=682 | -8.8 (80.05)
  LDH, Year 1 Week 48, n=692: number analyzed (Participants) | 692
  LDH, Year 1 Week 48, n=692 | -7.3 (81.32)
  LDH, Year 2 Week 24, n=641: number analyzed (Participants) | 641
  LDH, Year 2 Week 24, n=641 | -9.4 (85.83)
  LDH, Year 2 Week 48, n=592: number analyzed (Participants) | 592
  LDH, Year 2 Week 48, n=592 | -9.6 (95.52)
  LDH, Year 3 Week 24, n=532: number analyzed (Participants) | 532
  LDH, Year 3 Week 24, n=532 | -11.8 (93.90)
  LDH, Year 3 Week 48, n=486: number analyzed (Participants) | 486
  LDH, Year 3 Week 48, n=486 | -15.1 (94.65)
  LDH, Year 4 Week 24, n=438: number analyzed (Participants) | 438
  LDH, Year 4 Week 24, n=438 | -16.5 (99.93)
  LDH, Year 4 Week 48, n=418: number analyzed (Participants) | 418
  LDH, Year 4 Week 48, n=418 | -16.9 (102.11)
  LDH, Year 5 Week 24, n=393: number analyzed (Participants) | 393
  LDH, Year 5 Week 24, n=393 | -17.5 (106.45)
  LDH, Year 5 Week 48, n=362: number analyzed (Participants) | 362
  LDH, Year 5 Week 48, n=362 | -19.8 (108.33)
  LDH, Year 6 Week 24, n=303: number analyzed (Participants) | 303
  LDH, Year 6 Week 24, n=303 | -21.7 (115.77)
  LDH, Year 6 Week 48, n=284: number analyzed (Participants) | 284
  LDH, Year 6 Week 48, n=284 | -21.3 (122.62)
  LDH, Year 7 Week 24, n=182: number analyzed (Participants) | 182
  LDH, Year 7 Week 24, n=182 | -15.2 (44.05)
  LDH, Year 7 Week 48, n=130: number analyzed (Participants) | 130
  LDH, Year 7 Week 48, n=130 | -16.3 (42.51)
  LDH, Year 8 Week 24, n=52: number analyzed (Participants) | 52
  LDH, Year 8 Week 24, n=52 | -14.3 (40.14)
  LDH, Year 8 Week 48, n=13: number analyzed (Participants) | 13
  LDH, Year 8 Week 48, n=13 | -31.5 (53.04)
  LDH, Year 9 Week 24, n=6: number analyzed (Participants) | 6
  LDH, Year 9 Week 24, n=6 | -27.2 (32.64)
  LDH, Year 9 Week 48, n=1: number analyzed (Participants) | 1
  LDH, Year 9 Week 48, n=1 | -65.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  LDH, Exit, n=624: number analyzed (Participants) | 624
  LDH, Exit, n=624 | -13.1 (90.39)
  LDH, 8 Week follow-up, n=538: number analyzed (Participants) | 538
  LDH, 8 Week follow-up, n=538 | -12.7 (95.65)

16. Primary Outcome: Change From Baseline in Bilirubin (Bili) Levels
Description: Liver function parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 liver function parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Bili were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
µmol/L
  Year 1 Week 4, n=707: number analyzed (Participants) | 707
  Year 1 Week 4, n=707 | 0.142 (2.8398)
  Year 1 Week 12, n=705: number analyzed (Participants) | 705
  Year 1 Week 12, n=705 | 0.008 (2.6383)
  Year 1 Week 24, n=703: number analyzed (Participants) | 703
  Year 1 Week 24, n=703 | 0.217 (3.1280)
  Year 1 Week 36, n=684: number analyzed (Participants) | 684
  Year 1 Week 36, n=684 | 0.173 (2.7566)
  Year 1 Week 48, n=693: number analyzed (Participants) | 693
  Year 1 Week 48, n=693 | 0.367 (2.8441)
  Year 2 Week 24, n=643: number analyzed (Participants) | 643
  Year 2 Week 24, n=643 | 0.488 (2.9346)
  Year 2 Week 48, n=598: number analyzed (Participants) | 598
  Year 2 Week 48, n=598 | 0.540 (3.2181)
  Year 3 Week 24, n=535: number analyzed (Participants) | 535
  Year 3 Week 24, n=535 | 0.606 (3.1612)
  Year 3 Week 48, n=488: number analyzed (Participants) | 488
  Year 3 Week 48, n=488 | 0.637 (3.2474)
  Year 4 Week 24, n=439: number analyzed (Participants) | 439
  Year 4 Week 24, n=439 | 0.548 (2.9773)
  Year 4 Week 48, n=421: number analyzed (Participants) | 421
  Year 4 Week 48, n=421 | 0.629 (3.4680)
  Year 5 Week 24, n=393: number analyzed (Participants) | 393
  Year 5 Week 24, n=393 | 0.410 (2.6931)
  Year 5 Week 48, n=362: number analyzed (Participants) | 362
  Year 5 Week 48, n=362 | 0.788 (3.1324)
  Year 6 Week 24, n=304: number analyzed (Participants) | 304
  Year 6 Week 24, n=304 | 0.801 (2.9946)
  Year 6 Week 48, n=285: number analyzed (Participants) | 285
  Year 6 Week 48, n=285 | 0.638 (3.0669)
  Year 7 Week 24, n=183: number analyzed (Participants) | 183
  Year 7 Week 24, n=183 | 0.938 (2.8158)
  Year 7 Week 48, n=130: number analyzed (Participants) | 130
  Year 7 Week 48, n=130 | 1.129 (3.0314)
  Year 8 Week 24, n=52: number analyzed (Participants) | 52
  Year 8 Week 24, n=52 | 1.280 (3.0707)
  Year 8 Week 48, n=13: number analyzed (Participants) | 13
  Year 8 Week 48, n=13 | 0.768 (3.0434)
  Year 9 Week 24, n=6: number analyzed (Participants) | 6
  Year 9 Week 24, n=6 | 0.028 (2.0182)
  Year 9 Week 48, n=1: number analyzed (Participants) | 1
  Year 9 Week 48, n=1 | -2.870 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Exit, n=624: number analyzed (Participants) | 624
  Exit, n=624 | 0.573 (3.3274)
  8 Week follow-up, n=539: number analyzed (Participants) | 539
  8 Week follow-up, n=539 | 0.572 (3.1052)

17. Primary Outcome: Change From Baseline in Immunoglobulin G (IgG) Levels
Description: Immunoglobulin (Ig) parameters were assessed at Baseline, Week 4,12,24,36, and 48 during Year 1. From Year 2-9 Ig parameters were assessed at Week 24 and 48 ; Exit visit and at follow-up (up to 8 weeks post infusion). Change from Baseline in Ig G were summarized. The Baseline is defined as For Year 1, Day 0 values for MITT participants who were treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants who were treated with belimumab in the parent study. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 9 years
Population: MITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
g/L
  Year 1 Week 12, n=213: number analyzed (Participants) | 213
  Year 1 Week 12, n=213 | -1.571 (2.2970)
  Year 1 Week 24, n=709: number analyzed (Participants) | 709
  Year 1 Week 24, n=709 | -1.963 (2.7334)
  Year 1 Week 48, n=695: number analyzed (Participants) | 695
  Year 1 Week 48, n=695 | -2.507 (3.1054)
  Year 2 Week 24, n=482: number analyzed (Participants) | 482
  Year 2 Week 24, n=482 | -3.058 (3.6147)
  Year 2 Week 48, n=605: number analyzed (Participants) | 605
  Year 2 Week 48, n=605 | -3.232 (3.7414)
  Year 3 Week 24, n=143: number analyzed (Participants) | 143
  Year 3 Week 24, n=143 | -3.453 (3.7073)
  Year 3 Week 48, n=405: number analyzed (Participants) | 405
  Year 3 Week 48, n=405 | -3.791 (4.0450)
  Year 4 Week 24, n=146: number analyzed (Participants) | 146
  Year 4 Week 24, n=146 | -3.839 (4.1411)
  Year 4 Week 48, n=362: number analyzed (Participants) | 362
  Year 4 Week 48, n=362 | -3.794 (3.8780)
  Year 5 Week 24, n=111: number analyzed (Participants) | 111
  Year 5 Week 24, n=111 | -4.356 (3.6399)
  Year 5 Week 48, n=322: number analyzed (Participants) | 322
  Year 5 Week 48, n=322 | -4.323 (4.0169)
  Year 6 Week 24, n=71: number analyzed (Participants) | 71
  Year 6 Week 24, n=71 | -5.111 (3.8846)
  Year 6 Week 48, n=268: number analyzed (Participants) | 268
  Year 6 Week 48, n=268 | -4.697 (3.9599)
  Year 7 Week 24, n=50: number analyzed (Participants) | 50
  Year 7 Week 24, n=50 | -4.803 (3.5908)
  Year 7 Week 48, n=115: number analyzed (Participants) | 115
  Year 7 Week 48, n=115 | -4.982 (4.0769)
  Year 8 Week 24, n=18: number analyzed (Participants) | 18
  Year 8 Week 24, n=18 | -6.016 (3.8450)
  Year 8 Week 48, n=12: number analyzed (Participants) | 12
  Year 8 Week 48, n=12 | -5.520 (5.1564)
  Year 9 Week 48, n=1: number analyzed (Participants) | 1
  Year 9 Week 48, n=1 | 0.710 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Exit, n=627: number analyzed (Participants) | 627
  Exit, n=627 | -4.138 (4.0025)
  8 Week Follow up, n=543: number analyzed (Participants) | 543
  8 Week Follow up, n=543 | -4.325 (4.0246)

18. Primary Outcome: Number of Participants With Immunogenic Response by Year
Description: Immunogenic response was analyzed using serum samples for anti-belimumab antibody measurements in MITT population. Categories of response are Negative, Transient Positive (+) means single + response that does not occur at the final assessment, and Persistent + means + response that occurs at least 2 consecutive assessments or a single result at the final assessment. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Participants
  Year 0-1 Negative, n=717: number analyzed (Participants) | 717
  Year 0-1 Negative, n=717 | 707
  Year 1-2 Negative, n=684: number analyzed (Participants) | 684
  Year 1-2 Negative, n=684 | 656
  Year 2-3 Negative, n=590: number analyzed (Participants) | 590
  Year 2-3 Negative, n=590 | 577
  Year 3-4, Negative, n=502: number analyzed (Participants) | 502
  Year 3-4, Negative, n=502 | 498
  Year 4-5 Negative, n=432: number analyzed (Participants) | 432
  Year 4-5 Negative, n=432 | 432
  Year 5-6 Negative, n=336: number analyzed (Participants) | 336
  Year 5-6 Negative, n=336 | 336
  Year 6-7 Negative, n=212: number analyzed (Participants) | 212
  Year 6-7 Negative, n=212 | 212
  Year 7-8 Negative, n=64: number analyzed (Participants) | 64
  Year 7-8 Negative, n=64 | 64
  Year 8 plus Negative, n=6: number analyzed (Participants) | 6
  Year 8 plus Negative, n=6 | 6
  Year 0-1 Transient +, n=717: number analyzed (Participants) | 717
  Year 0-1 Transient +, n=717 | 10
  Year 1-2 Transient + n=684: number analyzed (Participants) | 684
  Year 1-2 Transient + n=684 | 18
  Year 2-3 Transient +, n=590: number analyzed (Participants) | 590
  Year 2-3 Transient +, n=590 | 9
  Year 3-4 Transient +, n=502: number analyzed (Participants) | 502
  Year 3-4 Transient +, n=502 | 4
  Year 4-5 Transient +, n=432: number analyzed (Participants) | 432
  Year 4-5 Transient +, n=432 | 0
  Year 5-6 Transient +, n=336: number analyzed (Participants) | 336
  Year 5-6 Transient +, n=336 | 0
  Year 6-7 Transient +, n=212: number analyzed (Participants) | 212
  Year 6-7 Transient +, n=212 | 0
  Year 7-8 Transient +, n=64: number analyzed (Participants) | 64
  Year 7-8 Transient +, n=64 | 0
  Year 8 plus Transient +, n=6: number analyzed (Participants) | 6
  Year 8 plus Transient +, n=6 | 0
  Year 0-1 Persistent+,n=717: number analyzed (Participants) | 717
  Year 0-1 Persistent+,n=717 | 0
  Year 1-2 Persistent+,n=684: number analyzed (Participants) | 684
  Year 1-2 Persistent+,n=684 | 10
  Year 2-3 Persistent+,n=590: number analyzed (Participants) | 590
  Year 2-3 Persistent+,n=590 | 3
  Year 3-4 Persistent+,n=502: number analyzed (Participants) | 502
  Year 3-4 Persistent+,n=502 | 0
  Year 4-5 Persistent+,n=432: number analyzed (Participants) | 432
  Year 4-5 Persistent+,n=432 | 0
  Year 5-6 Persistent+,n=336: number analyzed (Participants) | 336
  Year 5-6 Persistent+,n=336 | 0
  Year 6-7 Persistent+,n=212: number analyzed (Participants) | 212
  Year 6-7 Persistent+,n=212 | 0
  Year 7-8 Persistent+,n=64: number analyzed (Participants) | 64
  Year 7-8 Persistent+,n=64 | 0
  Year 8 plus Persistent+,n=6: number analyzed (Participants) | 6
  Year 8 plus Persistent+,n=6 | 0
  Year 0-1 Unknown, n=717: number analyzed (Participants) | 717
  Year 0-1 Unknown, n=717 | 0
  Year 1-2 Unknown, n=684: number analyzed (Participants) | 684
  Year 1-2 Unknown, n=684 | 0
  Year 2-3 Unknown, n=590: number analyzed (Participants) | 590
  Year 2-3 Unknown, n=590 | 1
  Year 3-4 Unknown, n=502: number analyzed (Participants) | 502
  Year 3-4 Unknown, n=502 | 0
  Year 4-5 Unknown, n=432: number analyzed (Participants) | 432
  Year 4-5 Unknown, n=432 | 0
  Year 5-6 Unknown, n=336: number analyzed (Participants) | 336
  Year 5-6 Unknown, n=336 | 0
  Year 6-7 Unknown, n=212: number analyzed (Participants) | 212
  Year 6-7 Unknown, n=212 | 0
  Year 7-8 Unknown, n=64: number analyzed (Participants) | 64
  Year 7-8 Unknown, n=64 | 0
  Year 8 plus Unknown, n=6: number analyzed (Participants) | 6
  Year 8 plus Unknown, n=6 | 0

19. Primary Outcome: Number of Participants With IgG Values Below the Lower Limit of Normal by Year
Description: Blood samples were collected to evaluate IgG levels at Baseline and at Weeks 12, 24 and 48 during Year 1. From Year 2-9, IgG was evaluated at Week 24 and 48 ; Exit visit and at follow-up visit (up to 8 weeks post last infusion). Number of participants with IgG immunoglobulin values below the LLN at each one year interval are presented. Baseline includes Extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with Belimumab in the parent study. If a participant had more than one response within a year, then the last response within the year interval (usually the Week 48 assessment) was summarized. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Participants
  Baseline, n=735 | 6
  Any Time Post Baseline, n=735 | 64
  Year 0-1, n=735 | 22
  Year 1-2, n=701: number analyzed (Participants) | 701
  Year 1-2, n=701 | 24
  Year 2-3, n=620: number analyzed (Participants) | 620
  Year 2-3, n=620 | 22
  Year 3-4, n=514: number analyzed (Participants) | 514
  Year 3-4, n=514 | 19
  Year 4-5, n=442: number analyzed (Participants) | 442
  Year 4-5, n=442 | 15
  Year 5-6, n=345: number analyzed (Participants) | 345
  Year 5-6, n=345 | 10
  Year 6-7, n=219: number analyzed (Participants) | 219
  Year 6-7, n=219 | 8
  Year 7-8, n=65: number analyzed (Participants) | 65
  Year 7-8, n=65 | 2
  More than 8 Years, n=6: number analyzed (Participants) | 6
  More than 8 Years, n=6 | 0

20. Primary Outcome: Number of Participants With Shifts From Baseline in Prednisone and Other Steroids Dose by Visit
Description: Participants who had improving SLE disease activity for at least 8 weeks, at the investigator's discretion, the steroid dose was reduced by reduction to 7.5 mg/day. If the participant continued to have stable or improving disease activity after 4 weeks on a reduced dose, then the investigator considered reducing the dose again. Baseline includes extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with Belimumab in the parent study. Number of participants with shifts from Baseline total daily dose category by visit is summarized.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Participants
Groups:
- Participants With no Prednisone and Other Steroids at Baseline: Participants were not receiving prednisone and other steroids at Baseline.
- Participants With Baseline Daily Dose of >0 to <=7.5 mg: Participants were receiving a daily dose of >0 to <=7.5 mg of prednisone and other steroids at Baseline.
- Participants With Baseline Daily Dose of >7.5 to <=40 mg: Participants were receiving a daily dose of >7.5 to <=40 mg of prednisone and other steroids at Baseline.
- Participants With Baseline Daily Dose of >40 mg: Participants were receiving a daily dose of >40 mg of prednisone and other steroids at Baseline.
Arm/Group | Participants With no Prednisone and Other Steroids at Baseline | Participants With Baseline Daily Dose of >0 to <=7.5 mg | Participants With Baseline Daily Dose of >7.5 to <=40 mg | Participants With Baseline Daily Dose of >40 mg
Number analyzed (Participants) | 43 | 227 | 462 | 1
Participants
  Total daily dose=0, Year 1, Week 24 | 40 | 5 | 1 | 0
  Total daily dose >0 to <=7.5, Year 1, Week 24 | 1 | 194 | 71 | 0
  Total daily dose >7.5 to <=40, Year 1, Week 24 | 2 | 18 | 376 | 1
  Total daily dose >40, Year 1, Week 24 | 0 | 0 | 1 | 0
  Total daily dose=0, Year 1, Week 48 | 40 | 13 | 13 | 0
  Total daily dose >0 to <=7.5, Year 1, Week 48 | 2 | 180 | 123 | 0
  Total daily dose >7.5 to <=40, Year 1, Week 48 | 0 | 19 | 301 | 1
  Total daily dose >40, Year 1, Week 48 | 1 | 0 | 4 | 0
  Total daily dose=0, Year 2, Week 24 | 39 | 19 | 20 | 0
  Total daily dose >0 to <=7.5, Year 2, Week 24 | 3 | 157 | 145 | 0
  Total daily dose >7.5 to <=40, Year 2, Week 24 | 0 | 25 | 237 | 1
  Total daily dose >40, Year 2, Week 24 | 0 | 0 | 5 | 0
  Total daily dose=0, Year 2, Week 48 | 36 | 24 | 21 | 0
  Total daily dose >0 to <=7.5, Year 2, Week 48 | 1 | 143 | 163 | 0
  Total daily dose >7.5 to <=40, Year 2, Week 48 | 1 | 26 | 195 | 1
  Total daily dose >40, Year 2, Week 48 | 0 | 0 | 1 | 0
  Total daily dose=0, Year 3, Week 24 | 33 | 19 | 25 | 0
  Total daily dose >0 to <=7.5, Year 3, Week 24 | 3 | 130 | 159 | 0
  Total daily dose >7.5 to <=40, Year 3, Week 24 | 1 | 27 | 157 | 1
  Total daily dose >40, Year 3, Week 24 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 3, Week 48 | 31 | 20 | 30 | 0
  Total daily dose >0 to <=7.5, Year 3, Week 48 | 3 | 122 | 127 | 0
  Total daily dose >7.5 to <=40, Year 3, Week 48 | 0 | 23 | 145 | 1
  Total daily dose >40, Year 3, Week 48 | 0 | 0 | 2 | 0
  Total daily dose=0, Year 4, Week 24 | 28 | 17 | 34 | 0
  Total daily dose >0 to <=7.5, Year 4, Week 24 | 3 | 110 | 134 | 0
  Total daily dose >7.5 to <=40, Year 4, Week 24 | 2 | 23 | 120 | 1
  Total daily dose >40, Year 4, Week 24 | 0 | 0 | 2 | 0
  Total daily dose=0, Year 4, Week 48 | 22 | 18 | 40 | 0
  Total daily dose >0 to <=7.5, Year 4, Week 48 | 3 | 100 | 129 | 1
  Total daily dose >7.5 to <=40, Year 4, Week 48 | 1 | 16 | 108 | 0
  Total daily dose >40, Year 4, Week 48 | 0 | 1 | 0 | 0
  Total daily dose=0, Year 5, Week 24 | 19 | 28 | 33 | 0
  Total daily dose >0 to <=7.5, Year 5, Week 24 | 3 | 84 | 124 | 1
  Total daily dose >7.5 to <=40, Year 5, Week 24 | 1 | 16 | 99 | 0
  Total daily dose >40, Year 5, Week 24 | 0 | 0 | 2 | 0
  Total daily dose=0, Year 5, Week 48 | 17 | 26 | 34 | 0
  Total daily dose >0 to <=7.5, Year 5, Week 48 | 1 | 75 | 119 | 1
  Total daily dose >7.5 to <=40, Year 5, Week 48 | 1 | 13 | 85 | 0
  Total daily dose >40, Year 5, Week 48 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 6, Week 24 | 10 | 25 | 33 | 0
  Total daily dose >0 to <=7.5, Year 6, Week 24 | 2 | 62 | 99 | 1
  Total daily dose >7.5 to <=40, Year 6, Week 24 | 0 | 10 | 76 | 0
  Total daily dose >40, Year 6, Week 24 | 0 | 0 | 2 | 0
  Total daily dose=0, Year 6, Week 48 | 10 | 24 | 35 | 0
  Total daily dose >0 to <=7.5, Year 6, Week 48 | 1 | 54 | 90 | 1
  Total daily dose >7.5 to <=40, Year 6, Week 48 | 0 | 11 | 68 | 0
  Total daily dose >40, Year 6, Week 48 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 7, Week 24 | 4 | 10 | 29 | 0
  Total daily dose >0 to <=7.5, Year 7, Week 24 | 0 | 41 | 64 | 1
  Total daily dose >7.5 to <=40, Year 7, Week 24 | 1 | 3 | 40 | 0
  Total daily dose >40, Year 7, Week 24 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 7, Week 48 | 4 | 3 | 24 | 0
  Total daily dose >0 to <=7.5, Year 7, Week 48 | 0 | 32 | 34 | 1
  Total daily dose >7.5 to <=40, Year 7, Week 48 | 0 | 6 | 29 | 0
  Total daily dose >40, Year 7, Week 48 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 8, Week 24 | 2 | 1 | 8 | 0
  Total daily dose >0 to <=7.5, Year 8, Week 24 | 0 | 13 | 15 | 1
  Total daily dose >7.5 to <=40, Year 8, Week 24 | 0 | 2 | 11 | 0
  Total daily dose >40, Year 8, Week 24 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 8, Week 48 | 1 | 0 | 5 | 0
  Total daily dose >0 to <=7.5, Year 8, Week 48 | 0 | 3 | 6 | 0
  Total daily dose >7.5 to <=40, Year 8, Week 48 | 0 | 2 | 1 | 0
  Total daily dose >40, Year 8, Week 48 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 9, Week 24 | 0 | 0 | 1 | 0
  Total daily dose >0 to <=7.5, Year 9, Week 24 | 0 | 1 | 3 | 0
  Total daily dose >7.5 to <=40, Year 9, Week 24 | 0 | 1 | 0 | 0
  Total daily dose >40, Year 9, Week 24 | 0 | 0 | 0 | 0
  Total daily dose=0, Year 9, Week 48 | 0 | 0 | 0 | 0
  Total daily dose >0 to <=7.5, Year 9, Week 48 | 0 | 1 | 4 | 0
  Total daily dose >7.5 to <=40, Year 9, Week 48 | 0 | 1 | 0 | 0
  Total daily dose >40, Year 9, Week 48 | 0 | 0 | 0 | 0

21. Primary Outcome: Number of Participants With Any SLICC/ ACR Damage Index Worsening (Change > 0) From Baseline by Visit
Description: The SLICC/ACR Damage Index was assessed every 48 weeks and at the exit visit as a measure of disease activity. It was developed to assess the accumulated damage since the onset of the disease. The number of participants with worsening in their SLICC/ACR Damage Index score compared with Baseline have been presented. Worsening was defined as a change in score (post-Baseline visit score - Baseline score) > 0. Baseline includes extension Year 1 Day 0 values for MITT participants treated with placebo in the parent study, and the last pre-treatment value in the parent study for MITT participants treated with Belimumab in the parent study. For years in which a participant was withdrawn from the study, the exit visit assessment was used in place of the Week 48 assessment for the year. This value was not carried forward through later years. Only those participants available at the specified time points (represented by n=X in the category titles) were analyzed.
Time Frame: Up to 9 years
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Belimumab 10mg/kg IV
Number analyzed (Participants) | 735
Participants
  Year 1,Week 48, n=716: number analyzed (Participants) | 716
  Year 1,Week 48, n=716 | 39
  Year 2,Week 48, n=667: number analyzed (Participants) | 667
  Year 2,Week 48, n=667 | 50
  Year 3,Week 48, n=580: number analyzed (Participants) | 580
  Year 3,Week 48, n=580 | 56
  Year 4,Week 48, n=488: number analyzed (Participants) | 488
  Year 4,Week 48, n=488 | 57
  Year 5,Week 48, n=423: number analyzed (Participants) | 423
  Year 5,Week 48, n=423 | 51
  Year 6,Week 48, n=330: number analyzed (Participants) | 330
  Year 6,Week 48, n=330 | 41
  Year 7,Week 48, n=213: number analyzed (Participants) | 213
  Year 7,Week 48, n=213 | 28
  Year 8,Week 48, n=65: number analyzed (Participants) | 65
  Year 8,Week 48, n=65 | 8
  Year 9,Week 48, n=6: number analyzed (Participants) | 6
  Year 9,Week 48, n=6 | 0

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious adverse events (AEs) were collected from the start of investigational product and until 8 Weeks after the last infusion of trial medication (Approximately 8 years plus)
Description: The MITT consisted of all randomized participants who received at least one dose of trial medication.
Arm/Group | Belimumab 10mg/kg IV
All-Cause Mortality (participants affected / at risk) | 11/735
Serious Adverse Events (participants affected / at risk) | 231/735
Other Adverse Events (participants affected / at risk) | 614/735
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 10mg/kg IV (N=735)
Pneumonia bacterial (Infections and infestations) | 14 (16)
Cellulitis (Infections and infestations) | 12 (14)
Lupus nephritis (Renal and urinary disorders) | 12 (14)
Pyrexia (General disorders) | 9 (10)
Urinary tract infection (Infections and infestations) | 9 (9)
Urinary tract infection bacterial (Infections and infestations) | 9 (11)
Leukopenia (Blood and lymphatic system disorders) | 8 (9)
Pneumonia (Infections and infestations) | 8 (8)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Appendicitis (Infections and infestations) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Cholelithiasis (Hepatobiliary disorders) | 5 (5)
Gastritis (Gastrointestinal disorders) | 5 (5)
Gastroenteritis (Infections and infestations) | 5 (5)
Herpes zoster (Infections and infestations) | 5 (5)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 (10)
Raynaud's phenomenon (Vascular disorders) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Lupus vasculitis (Vascular disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bacterial pyelonephritis (Infections and infestations) | 3 (3)
Bacterial sepsis (Infections and infestations) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Septic shock (Infections and infestations) | 3 (4)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 3 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Abscess soft tissue (Infections and infestations) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
Acute sinusitis (Infections and infestations) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Bronchitis bacterial (Infections and infestations) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (4)
Diarrhoea infectious (Infections and infestations) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Escherichia infection (Infections and infestations) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Soft tissue infection (Infections and infestations) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 2 (2)
Suicide attempt (Psychiatric disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Vasculitis (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound infection bacterial (Infections and infestations) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abscess of salivary gland (Infections and infestations) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Amoebic dysentery (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Aortic valve sclerosis (Cardiac disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Complication associated with device (General disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Cutaneous tuberculosis (Infections and infestations) | 1 (1)
Cyst (General disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (2)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1)
Gallbladder non-functioning (Hepatobiliary disorders) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Gastrointestinal fungal infection (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1)
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Joint tuberculosis (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (3)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1)
Latent tuberculosis (Infections and infestations) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lupus enteritis (Gastrointestinal disorders) | 1 (2)
Lupus hepatitis (Hepatobiliary disorders) | 1 (1)
Lupus myocarditis (Cardiac disorders) | 1 (1)
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Maculopathy (Eye disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (2)
Migraine (Nervous system disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropsychiatric lupus (Nervous system disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 1 (1)
Parovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pericarditis lupus (Cardiac disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin candida (Infections and infestations) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab 10mg/kg IV (N=735)
Headache (Nervous system disorders) | 205 (407)
Nasopharyngitis (Infections and infestations) | 155 (396)
Diarrhoea (Gastrointestinal disorders) | 143 (235)
Arthralgia (Musculoskeletal and connective tissue disorders) | 134 (217)
Influenza (Infections and infestations) | 132 (274)
Cough (Respiratory, thoracic and mediastinal disorders) | 120 (176)
Back pain (Musculoskeletal and connective tissue disorders) | 102 (141)
Urinary tract infection bacterial (Infections and infestations) | 87 (163)
Viral upper respiratory tract infection (Infections and infestations) | 84 (196)
Upper respiratory tract infection (Infections and infestations) | 82 (151)
Pyrexia (General disorders) | 73 (92)
Urinary tract infection (Infections and infestations) | 68 (99)
Hypertension (Vascular disorders) | 67 (111)
Myalgia (Musculoskeletal and connective tissue disorders) | 64 (77)
Nausea (Gastrointestinal disorders) | 64 (97)
Dizziness (Nervous system disorders) | 61 (82)
Abdominal pain (Gastrointestinal disorders) | 60 (78)
Abdominal pain upper (Gastrointestinal disorders) | 60 (80)
Fatigue (General disorders) | 56 (61)
Rash (Skin and subcutaneous tissue disorders) | 56 (77)
Herpes zoster (Infections and infestations) | 55 (56)
Insomnia (Psychiatric disorders) | 55 (64)
Upper respiratory tract infection bacterial (Infections and infestations) | 54 (108)
Gastritis (Gastrointestinal disorders) | 52 (59)
Vomiting (Gastrointestinal disorders) | 50 (70)
Depression (Psychiatric disorders) | 49 (57)
Gastroenteritis (Infections and infestations) | 49 (59)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 (73)
Alopecia (Skin and subcutaneous tissue disorders) | 48 (62)
Bronchitis bacterial (Infections and infestations) | 48 (81)
Oedema peripheral (General disorders) | 47 (56)
Bronchitis (Infections and infestations) | 46 (64)
Anaemia (Blood and lymphatic system disorders) | 45 (56)
Oral herpes (Infections and infestations) | 45 (89)
Pruritus (Skin and subcutaneous tissue disorders) | 44 (55)
Dyspepsia (Gastrointestinal disorders) | 39 (50)
Hypotension (Vascular disorders) | 39 (192)
Pharyngitis bacterial (Infections and infestations) | 39 (85)
Non-cardiac chest pain (General disorders) | 38 (41)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 37 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.